CLINICAL TRIAL: NCT00932451
Title: Phase 2, Open-label Single Arm Study Of The Efficacy And Safety Of Pf-02341066 In Patients With Advanced Non-small Cell Lung Cancer (Nsclc) Harboring A Translocation Or Inversion Involving The Anaplastic Lymphoma Kinase (Alk) Gene Locus
Brief Title: An Investigational Drug, PF-02341066, Is Being Studied In Patients With Advanced Non-Small Cell Lung Cancer With A Specific Gene Profile Involving The Anaplastic Lymphoma Kinase (ALK) Gene
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: A8081005; 2009-012504-13 (EudraCT Number)
Record Dates: First submitted 2009-06-30; First posted 2009-07-03 (Estimated); Results first posted 2016-06-09 (Estimated); Last update posted 2017-01-13 (Estimated); Status verified 2016-11

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Lung Neoplasms ALK gene Crizotinib
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Crizotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PF-0231066 (Experimental)
  Interventions: Drug: PF-02341066

INTERVENTIONS:
Drug: PF-02341066 — PF-02341066, 250 mg BID, will be administered orally on a continuous schedule

SUMMARY:
This is a Phase 2 trial that will evaluate the safety and efficacy of PF-02341066 in patients with advanced non-small cell lung cancer with a specific gene profile involving the ALK gene. This trial will also allow patients from a Phase 3 trial who received standard of care chemotherapy (Study A8081007) to receive PF-02341066.

ELIGIBILITY:
Inclusion Criteria:

* histologically or cytologically proven diagnosis of non-small cell lung cancer
* positive for the ALK fusion gene (test provided by either a central laboratory. Local laboratory may be used for certain cases)
* may have received pemetrexed or docetaxel from previous Phase 3 trial (A8081007) and discontinued treatment due to Response Evaluation Criterion in Solid Tumors (RECIST)-defined progression. or, once the primary endpoint of Study A8081007 has been analyzed and the results made available, at any time without RECIST-defined progression.
* Tumors can be measurable or non measurable

Exclusion Criteria:

* prior treatment with PF-02341066
* received no prior systemic treatment, chemotherapy or EGFR tyrosine kinase inhibitor, for advanced non-small cell lung cancer
* current enrollment in another therapeutic clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1069 (Actual)
Dates: Start 2010-01; Primary Completion 2015-03 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (275):
- United States (136):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Comprehensive Blood and Cancer Center, Bakersfield, California
  - Tower Cancer Research Foundation, Beverly Hills, California
  - Tower Hematology Oncology Medical Group, Beverly Hills, California
  - Moores UCSD Cancer Center, La Jolla, California
  - UCSD Medical Center - La Jolla, La Jolla, California
  - Drug Shipping Address: Ronald Reagen University of California-Los Angeles, Los Angeles, California
  - Ronald Reagen University of California-Los Angeles Medical Center, Los Angeles, California
  - UCLA Opthalmic Oncology Center, Los Angeles, California
  - University of California-Los Angeles, Los Angeles, California
  - University of California, Irvine-Medical Center, Orange, California
  - University of California, Irvine-Pharmacy, Orange, California
  - Stanford University-Cancer Center, Palo Alto, California
  - UC Davis Cancer Center, Sacramento, California
  - University of California Davis Medical Center, Sacramento, California
  - UCSD Medical Center - Hillcrest, San Diego, California
  - Santa Monica-UCLA Medical Center & Orthopaedic Hospital Clinical Laboratory, Santa Monica, California
  - UCLA Hematology Oncology-Santa Monica, Santa Monica, California
  - University of California-Los Angeles, Santa Monica, California
  - Redwood Regional Medical Group Inc, Santa Rosa, California
  - DRUG SHIPMENT: University of Colorado Cancer Center, Aurora, Colorado
  - Rocky Mountain Lions Eye Institute, Aurora, Colorado
  - University of Colorado Hospital, Aurora, Colorado
  - Kaiser Permanente Colorado - Franklin, Denver, Colorado
  - Kaiser Permanente Colorado - Rock Creek, Lafayette, Colorado
  - Smilow Cancer Center at Yale New Haven, Oncology Pharmacy, New Haven, Connecticut
  - Smilow Cancer Hospital at Yale New Haven, New Haven, Connecticut
  - Yale University, New Haven, Connecticut
  - Michael and Dianne Bienes Cancer Center, Holy Cross Hospital, Fort Lauderdale, Florida
  - Memorial Cancer Institute, Hollywood, Florida
  - Cancer Center of South Florida Foundation, Inc., Lake Worth, Florida
  - Memorial Cancer Center (West), Pembroke Pines, Florida
  - H Lee Moffitt Cancer Center & Research Institute, Tampa, Florida
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory Clinic, Atlanta, Georgia
  - Emory University Clinic, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia
  - Winship Cancer Institution, Atlanta, Georgia
  - Georgia Cancer Specialists - Administrative Annex, Atlanta, Georgia
  - MCG Health Cancer Center Pharmacy, Augusta, Georgia
  - MCG Health System Pharmacy (Drug Shipment Only), Augusta, Georgia
  - Medical College of Georgia, Augusta, Georgia
  - Georgia Cancer Specialists-Stemmer, Decatur, Georgia
  - Georgia Cancer Specialists-Macon, Macon, Georgia
  - Georgia Cancer Specialists-Kennestone, Marietta, Georgia
  - Georgia Cancer Specialists-Northside, Sandy Springs, Georgia
  - OnCare Hawaii, Inc., Honolulu, Hawaii
  - University of Hawaii - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - Hawaii Medical Center East, Honolulu, Hawaii
  - Rush University Medical Center, Chicago, Illinois
  - University of Chicago Medical Center (Attn: J Pi PharmD / A. Patel Pharm D), Chicago, Illinois
  - University of Chicago Medical Center, Chicago, Illinois
  - Ingalls Memorial Hospital (Drug Shipment Only), Harvey, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Monroe Medical Associates, Harvey, Illinois
  - Monroe Medical Associates, Tinley Park, Illinois
  - Indiana University Hospital Clarian Health, Indianapolis, Indiana
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Ship drug to: Investigational Drug Services, Indianapolis, Indiana
  - Wishard Memorial Hospital, Indianapolis, Indiana
  - Springmill Medical Clinic, Indianopolis, Indiana
  - Monroe Medical Associates, Munster, Indiana
  - The Community Hospital, Munster, Indiana
  - Johns Hopkins Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - The Harry and Jeanette Cancer Research Building, Baltimore, Maryland
  - National Institutes of Health National Cancer Institute, Bethesda, Maryland
  - Massachusette General Hospital, Boston, Massachusetts
  - Massachussetts General Hospital, Boston, Massachusetts
  - Beth Isreal Deaconess Medical Center, Pharmacy FD B18, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Beth Isreal Deaconess Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Institute/Pharmacy, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - Karmanos Cancer lnstitute at Farmington Hllls, Farmington Hills, Michigan
  - Siteman Cancer Center, City of Saint Peters, Missouri
  - Barnes-Jewish Hospital, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Dartmouth Hitchcock Medical Center/Mary Hitchcock Memorial Hospital, Lebanon, New Hampshire
  - University of New Mexico Eye Clinic, Albuquerque, New Mexico
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - NSLIJ Health System/Monter Cancer Center, Lake Success, New York
  - North Shore University Hospital, Manhasset, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - Memorial Sloan-Kettering Cancer Center: Rockefeller Outpatient Pavilion, New York, New York
  - Columbia University Medical Center, New York, New York
  - IP Shipment: CUMC Research Pharmacy, New York, New York
  - Memorial Sloan - Kettering Cancer Center, New York, New York
  - Department of Medicine MSG at SUNY HSC at Syracuse, INC., d/b/a University Physicians, Oneida, New York
  - Department of Medicine MSG at SUNY HSC at Syracuse, INC., d/b/a University Physicians, Oswego, New York
  - SUNY Upstate Medical University, Regional Oncology Center, Syracuse, New York
  - Department of Medicine MSG at SUNY HSC at Syracuse, INC., d/b/a University Physicians, Syracuse, New York
  - UNC Health Care, Chapel Hill, North Carolina
  - UNC Hospitals, The University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Presbyterian Hospital Cancer Center, Charlotte, North Carolina
  - Presbyterian Hospital Huntersville, Huntersville, North Carolina
  - Southern Oncology Specialists, Huntersville, North Carolina
  - Presbyterian Hospital Matthews, Matthews, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - The Ohio State University Hospital East, Columbus, Ohio
  - The Ohio State University Investigational Drug Services, Columbus, Ohio
  - The Ohio State University James Cancer Hospital and Solove Research Institute, Columbus, Ohio
  - James Care in Kenny, Columbus, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Penn State Milton S. Hershey Medical Center, Penn State Hershey Cancer Institute, Hershey, Pennsylvania
  - Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Penn Presbyterian Medical Center, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Vincent Armenio, MD, East Providence, Rhode Island
  - Pharma Resource, East Providence, Rhode Island
  - Medical University of South Carolina - Hollings Cancer Center, Charleston, South Carolina
  - Tennessee Oncology, PLLC, Dickson, Tennessee
  - Tennessee Oncology, PLLC, Franklin, Tennessee
  - Tennessee Oncology, PLLC, Gallatin, Tennessee
  - Tennessee Oncology, PLLC, Hermitage, Tennessee
  - Tennessee Oncology, PLLC, Lebanon, Tennessee
  - Tennessee Oncology, PLLC, Murfreesboro, Tennessee
  - Sarah Cannon Research Institute (Administration), Nashville, Tennessee
  - Sarah Cannon Research Institute (Pharmacy), Nashville, Tennessee
  - Tennessee Oncology, PLLC, Nashville, Tennessee
  - Vanderbilt Cancer Clinic, Nashville, Tennessee
  - The Vanderbilt Chemo Clinic, Nashville, Tennessee
  - Tennessee Oncology, PLLC, Smyrna, Tennessee
  - UT Southwestern Medical Center - Simmons Cancer Center Pharmacy, Dallas, Texas
  - University of Texas Southwestern Medical Center at Dallas, Dallas, Texas
  - University of Texas Southwestern University Hospital - Zale Lipshy, Dallas, Texas
  - UT Southwestern University Hospital - William P. Clements, Jr, Dallas, Texas
  - The University of Texas, Houston, Texas
  - Swedish Cancer Institute, Seattle, Washington
  - Seattle Cancer Care Alliance, Seattle, Washington
  - Lisa Nakatsu, RPh (Drug Shipment Address), Seattle, Washington
  - Swedish Medical Center, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
- Australia (4):
  - Chris O'Brien Lifehouse, Camperdown, New South Wales
  - Royal Adelaide Hospital, Department of Medical Oncology, Adelaide, South Australia
  - Peter MacCallum Cancer Centre, Division of Haematology and Medical Oncology, East Melbourne, Victoria
  - Department of Medical Oncology, Nedlands, Western Australia
- Brazil (9):
  - Nucleo de Oncologia da Bahia, Salvador, Estado de Bahia
  - Instituto Nacional do Câncer - INCA, Rio de Janeiro, Rio de Janeiro
  - Associacao Hospital de Caridade de Ijui, Ijuí, Rio Grande do Sul
  - Irmandade da Santa Casa de Misericordia de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Hospital Sao Lucas da PUCRS, Porto Alegre, Rio Grande do Sul
  - Fundacao Pio XII Hospital de Cancer de Barretos, Barretos, São Paulo
  - Fundacao Hospital Amaral Carvalho, Jaú, São Paulo
  - Instituto do Câncer do Estado de São Paulo Octavio Frias de Oliveira - ICESP, São Paulo, São Paulo
  - Fundacao Antonio Prudente, São Paulo, São Paulo
- Bulgaria (4):
  - UMHAT Tsaritsa Yoanna - ISUL, Sofia, Bulgaria
  - Spetsializirana Bolnitsa za Aktivno Lechenie po Onkologiya, Klinika po himioterapiya, Sofia, Bulgaria
  - MBAL Voennomeditsinska Academia, MMA HAT Sofia, Sofia
  - MDOZS "Dr. Marko Markov", Otdelenie po onkoterapiya i paliativni grizhi, Varna
- Canada (14):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Alberta Health Services, Holy Cross Site, Calgary, Alberta
  - Office of Dr. John McWhae, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - Dr. Georges-L. Dumont Regional Hospital, Moncton, New Brunswick
  - Dr. Leon Richard Oncology Centre, Moncton, New Brunswick
  - RSM Durham Regional Cancer Centre - Lakeridge Health Oshawa, Oshawa, Ontario
  - Dr. Dana Blakolmer and Associates, Oshawa, Ontario
  - The Ottawa Hospital Cancer Center, Ottawa, Ontario
  - Hopital Notre-Dame du Centre Hospitalier de l'Universite de Montreal (CHUM), Montreal, Quebec
  - Royal Victoria Hospital, Montreal, Quebec
  - Montreal General Hospital, Montreal, Quebec
  - Jewish General Hospsital, Montreal, Quebec
  - St. Mary's Hospital Center, Montreal, Quebec
- China (9):
  - SUN Yat-Sen University Cancer Center, Guangzhou, Guangdong
  - Nanjing Bayi Hospital, Nanjing, Jiangsu
  - Cancer Institute and Hospital Chinese Academy of Medical Sciences and PUMC, Internal 4 Department, Beijing
  - 307 Hospital of PLA, Beijing
  - Guangdong General Hospital, Guangzhou
  - Shanghai Chest Hospital/Department of Pulmonary Medicine, Shanghai
  - Shanghai Chest Hospital, Shanghai
  - Zhongshan Hospital Fudan University / Respiratory Department, Shanghai
  - Shanghai Pulmonary Hospital, Shanghai
- France (9):
  - Centre Francois Baclesse, Caen
  - Centre Georges-François Leclerc, Dijon
  - Hopital Albert Michallon, Grenoble
  - APHM - Hopital Nord / Service d'Oncologie Multidisciplinaire et Innovations Thérapeutiques, Marseille
  - Centre Antoine Lacassagne, Nice
  - Hospital Cochin, Paris
  - Hopital Tenon, Paris
  - Centre Rene Gauducheau / Service d'Oncologie Medicale, Saint-Herblain
  - Institut Gustave Roussy, Villejuif
- Germany (9):
  - Klinikum der Universitaet zu Koeln, Klinik I fuer Innere Medizin, Cologne
  - Universitaetsklinikum Carl-Gustav-Carus Dresden, Dresden
  - Westdeutsches Tumorzentrum, Universitaetsklinikum Essen, Innere Klinik - Tumorforschung, Essen
  - Krankenhaus Grosshansdorf, Zentrum fuer Pneumologie und Thoraxchirurgie, Großhansdorf
  - Ambulantes Krebszentrum Hamburg, Hamburg
  - Thoraxklinik Heidelberg gGmbH, Heidelberg
  - Klinikum der Universitaet Muenchen, Medizinische Klink - Innenstadt, Pneumologie, München
  - Pius-Hospital Oldenburg, Oldenburg
  - HSK Dr.- Horst-Schmidt-Kliniken, Wiesbaden
- Greece (3):
  - University General Hospital of Heraklion/ Department of Clinical Oncology, Heraklion, Crete
  - General Hospital of Thessaloniki Georgios Papanikolaou, Lung Cancer Neoplasia Research Department, Eksochi, Thessaloniki
  - General Hospital of Chest Diseases of Athens "Sotiria", Athens
- Hong Kong (3):
  - Division of Respiratory and Critical Care Medicine, Department of Medicine, Queen Mary Hospital, Pokfulam
  - Department of Clinical Oncology, Prince of Wales Hospital, Shatin, New Territories
  - Tuen Mun Hospital, Department of Clinical Oncology, Tuen Mun, New Territories
- Hungary (6):
  - Orszagos Koranyi TBC es Pulmonologiai Intezet, VI. Bronchologia, Budapest
  - Semmelweis Egyetem Pulmonologia Intezet, Budapest
  - Debreceni Egyetem Orvos - es Egeszsegtudomanyi Centrum, Tudogyogyaszati Klinika, Debrecen
  - Veszprem Megyei Onkormanyzat Tudogyogyintezete, Farkasgyepű
  - Fejer Megyei Szent Gyorgy Korhaz, Pulmonologiai Osztaly, Székesfehérvár
  - Pest Megyei Tudogyogyintezet, III. Osztaly, Törökbálint
- Ireland (5):
  - Aseptic Compounding Unit, Dublin, Dublin
  - Department of Medical Oncology, Dublin, Dublin
  - Department of Medical Oncology, Galway, Ireland
  - Merlin Park Imaging Centre, Galway, Ireland
  - Pharmacy Aseptic Services Unit, Galway, Ireland
- Italy (14):
  - Divisione di Oncologia Medica, Ospedale San Giuseppe Moscati, Citta' Ospedaliera, Avellino
  - S.C. Oncologia Medica, Florence
  - Oncologia Medica A, Genova
  - Ospedale Versilia, Oncologia Medica, Lido Di Camaiore (LU)
  - Ospedale San Luca, Lucca
  - Dipartimento Oncologia Medica, UO Medicina 1Q A, Unita' Nuovi Farmaci e Terapie Innovative, Milan
  - Farmacia Istituto Europeo di Oncologia, Milan
  - Istituto Europeo di Oncologia, Milan
  - Ospedale Niguarda Ca' Granda Dipartimento Oncologico, SC Divisione di Oncologia Medica Falk, Milan
  - Nuovo Ospedale San Gerardo, Monza
  - Azienda Ospedaliera Universitaria San Luigi Gonzaga, Orbassano (TO)
  - SC Oncologia Medica, Ospedale Santa Maria della Misericordia, Azienda Ospedaliera di Perugia, Perugia
  - Unita' Operativa Complessa di Pneumologia Oncologica I, Padiglione Flaiani, Roma
  - Centro C.O.E.S., A.O. San Giovanni Battista Le Molinette, Torino
- Japan (10):
  - Aichi cancer center central hospital, Nagoya, Aichi-ken
  - National Hospital Organization Hokkaido Cancer Center, Sapporo, Hokkaido
  - Hyogo Cancer Center, Akashi, Hyōgo
  - Okayama University Hospital, Okayama, Okayama-ken
  - Kinki University Hospital, Osakasayama-shi, Osaka
  - Shizuoka Cancer Center, Sunto-gun, Shizuoka
  - National Cancer Center Hospital, Chuo-ku, Tokyo
  - National Kyushu Cancer Center/Department of Thoracic Oncology, Fukuoka
  - National Cancer Center Hospital East, Kashiwa
  - The Cancer Institute Hospital of JFCR, Tokyo
- Universitair Medisch Centrum Groningen, Groningen, Netherlands
- Poland (8):
  - Uniwersyteckie Centrum Kliniczne, Gdansk, Poland
  - Pracownia Optyczna Bozena Lawrynowicz Optyk Dyplomowany, Olsztyn, Poland
  - Ars Medica, Olsztyn, Poland
  - Wojewodzki Szpital Specjalistyczny w Olsztynie, Zaklad Medycyny Nuklearnej, Olsztyn, Poland
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Samodzielny Publiczny Zespol Gruzlicy i Chorob Pluc, Olsztyn
  - Oddzial Onkologii Klinicznej z Pododdzialem Dziennej Chemioterapii, Poznan
  - Zaklad Diagnostyki Obrazowej, Poznan
- Russia (5):
  - Republican Clinical Oncology Dispensary of the Ministry of Health of Tatarstan Republic, Kazan'
  - State Institution "National Cancer Research Center named after N.N. Blokhin' RAMS", Moscow
  - City Clinical Oncology Dispensary, Saint Petersburg
  - Saint-Petersburg State Medical University named after I.P.Pavlov of Roszdrav, Saint Petersburg
  - Research Institute of Pulmonology, Saint Petersburg
- South Korea (3):
  - National Cancer Center, Center for Lung Cancer, Gyeonggi-do
  - Seoul National University Hospital / Department of Internal Medicine, Seoul
  - Samsung Medical Center, Sungkyunkwan Univ School of Medicine, Seoul
- Spain (11):
  - Hospital Universitari Germans Trias I Pujol, Badalona, Barcelona
  - Hospital Del Mar, Barcelona, Barcelona
  - Hospital General Universitari Vall D´Hebron, Barcelona, Barcelona
  - Institut Catala D'Oncologia - Hospital Duran I Reynals, L'Hospitalet de Llobregat, Barcelona
  - Consorcio Hospitalario Parc Tauli, Sabadell, Barcelona
  - Hospital Universitario Marques de Valdecilla, Santander, Cantabria
  - Complexo Hospitalario Universitario A Coruña, A Coruña, Galicia
  - Hospital Universitario La Paz, Madrid, Madrid
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias
  - Hospital Universitario Virgen Del Rocio, Seville, Sevilla
  - Hospital de Navarra, Pamplona
- Karolinska Universitetssjukhuset, Onkologiska kliniken, Stockholm, Sweden
- Taiwan (3):
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Department of Internal Medicine, Taipei
  - Taipei Veterans General Hospital, Chest Department, Taipei
- United Kingdom (8):
  - Cancer and Haematology Centre,, Headington, Oxford
  - Royal Marsden Hospital, Sutton, Surrey
  - Nuffield Health Wessex Hospital, Eastleigh
  - Department of Oncology, London
  - Kings College London at Guy's Hospital, London
  - Royal Marsden Hospital, London
  - Christie Hospital NHS Trust, Department of Medical Oncology, Manchester
  - Somers Cancer Research Building, M824, Southampton

REFERENCES:
- [Derived] Camidge DR, Kim EE, Usari T, Polli A, Lewis I, Wilner KD. Renal Effects of Crizotinib in Patients With ALK-Positive Advanced NSCLC. J Thorac Oncol. 2019 Jun;14(6):1077-1085. doi: 10.1016/j.jtho.2019.02.015. Epub 2019 Feb 26. PMID 30822515
- [Derived] Blackhall F, Ross Camidge D, Shaw AT, Soria JC, Solomon BJ, Mok T, Hirsh V, Janne PA, Shi Y, Yang PC, Pas T, Hida T, Carpeno JC, Lanzalone S, Polli A, Iyer S, Reisman A, Wilner KD, Kim DW. Final results of the large-scale multinational trial PROFILE 1005: efficacy and safety of crizotinib in previously treated patients with advanced/metastatic ALK-positive non-small-cell lung cancer. ESMO Open. 2017 Aug 17;2(3):e000219. doi: 10.1136/esmoopen-2017-000219. eCollection 2017. PMID 29209525
- [Derived] Yoneda KY, Scranton JR, Cadogan MA, Tassell V, Nadanaciva S, Wilner KD, Stollenwerk NS. Interstitial Lung Disease Associated With Crizotinib in Patients With Advanced Non-Small Cell Lung Cancer: Independent Review of Four PROFILE Trials. Clin Lung Cancer. 2017 Sep;18(5):472-479. doi: 10.1016/j.cllc.2017.03.004. Epub 2017 Mar 14. PMID 28373069
- [Derived] Lin YT, Yu CJ, Yang JC, Shih JY. Anaplastic Lymphoma Kinase (ALK) Kinase Domain Mutation Following ALK Inhibitor(s) Failure in Advanced ALK Positive Non-Small-Cell Lung Cancer: Analysis and Literature Review. Clin Lung Cancer. 2016 Sep;17(5):e77-e94. doi: 10.1016/j.cllc.2016.03.005. Epub 2016 Mar 30. PMID 27130468
- [Derived] Costa DB, Shaw AT, Ou SH, Solomon BJ, Riely GJ, Ahn MJ, Zhou C, Shreeve SM, Selaru P, Polli A, Schnell P, Wilner KD, Wiltshire R, Camidge DR, Crino L. Clinical Experience With Crizotinib in Patients With Advanced ALK-Rearranged Non-Small-Cell Lung Cancer and Brain Metastases. J Clin Oncol. 2015 Jun 10;33(17):1881-8. doi: 10.1200/JCO.2014.59.0539. Epub 2015 Jan 26. PMID 25624436
- [Derived] Lin YT, Wang YF, Yang JC, Yu CJ, Wu SG, Shih JY, Yang PC. Development of renal cysts after crizotinib treatment in advanced ALK-positive non-small-cell lung cancer. J Thorac Oncol. 2014 Nov;9(11):1720-5. doi: 10.1097/JTO.0000000000000326. PMID 25436806
- [Derived] Ou SH. Crizotinib: a drug that crystallizes a unique molecular subset of non-small-cell lung cancer. Expert Rev Anticancer Ther. 2012 Feb;12(2):151-62. doi: 10.1586/era.11.186. PMID 22316363
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A8081005&StudyName=An%20Investigational%20Drug%2C%20PF-02341066%2C%20Is%20Being%20Studied%20In%20Patients%20With%20Advanced%20Non-Small%20Cell%20Lung%20Cancer%20With%20A%20Specific%20Gene%20Pro

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 1069 participants entered the study out of which 3 participants were withdrawn from the study before receiving study treatment because they were not eligible and were mistakenly entered into the interactive voice response system. Only 1066 participants received greater than or equal to 1 dose of crizotinib.
Pre-assignment Details: A total of 144 participants in study NCT00932893 were also enrolled in this study to receive treatment with crizotinib, including 143 participants randomized to the chemotherapy arm then crossed over in this study and 1 participant initially erroneously randomized in the crizotinib arm but not treated.
Groups:
- Crizotinib 250 mg BID: Participants were administered crizotinib at a starting dose of 250 mg orally, BID on a continuous dosing period as two 100-mg tablets and one 50-mg tablet at approximately 12 hours apart the same time each day.
Period: Overall Study
Arm/Group | Crizotinib 250 mg BID
Started | 1066
Completed | 244
Not Completed | 822
Not completed — Withdrawal by Subject | 69
Not completed — Lost to Follow-up | 22
Not completed — Death | 726
Not completed — Other reasons | 5

BASELINE CHARACTERISTICS:
Population: An Investigational Use Only (IUO) population (N=908) was all participants whose non-small cell lung cancer (NSCLC) was Fluorescent In-Situ Hybridization (FISH) ALK (Anaplastic Lymphoma Receptor Tyrosine Kinase) (+) by the central laboratory. A non-IUO population (N=158) was all partcipants whose NSCLC was ALK (+) by local assay testing.
Arm/Group | Crizotinib 250 mg BID
Number analyzed (Participants) | 1066
Age, Continuous [Mean (Standard Deviation); unit: Years] | 52.2 (12.33)
Age, Customized [Number; unit: Participants]
  < 65 years | 894
  >=65 years | 172
Gender [Count of Participants; unit: Participants]
  Female | 601
  Male | 465
Race/Ethnicity, Customized [Number; unit: participants]
  Chinese | 252
  Japanese | 81
  Korean | 144
  White | 532
  Black | 20
  Other | 19
  Other-Asian | 18

OUTCOME MEASURES:

1. Secondary Outcome: Duration of Response (DR)
Description: DR was defined as the time from the first documentation of objective tumor response (CR or PR) that was subsequently confirmed, to the first documentation of objective tumor progression or to death on study due to any cause, whichever occurred first. DR (in months) was calculated as (first date of PD or death - first date of CR or PR that was subsequently confirmed + 1)/30.4.
Time Frame: 6 years
Population: Response-evaluable populations: defined as participants in either the SA-ALK positive by IUO population or SA-ALK positive by non-IUO population, respectively, who had adequate baseline tumor assessment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Crizotinib 250 mg BID
Number analyzed (Participants) | 1066
Months
  ALK Positive by IUO, N=491 | 11.8 [10.4 to 12.8]
  ALK Positive by non-IUO only, N=64 | 9.5 [6.9 to 15.2]

2. Secondary Outcome: Time to Tumor Response (TTR)
Description: TTR was defined as the time (in weeks) from the date of Cycle 1 Day 1 dose to first documentation of objective tumor response (CR or PR) that was subsequently confirmed. For participants proceeding from PR to CR, the onset of PR was taken as the onset of response.
Time Frame: 6 years
Population: as for outcome 1
Measure: Median (Full Range); unit: Weeks
Arm/Group | Crizotinib 250 mg BID
Number analyzed (Participants) | 1066
Weeks
  ALK Positive by IUO (n=491) | 6.1 [2.7 to 164]
  ALK Positive by non-IUO only (n=64) | 6.3 [4.7 to 65.9]

3. Secondary Outcome: Disease Control Rate (DCR)
Description: DCR at 6 and 12 weeks was defined as the percentage of participants with a confirmed CR, confirmed PR, or SD (according to RECIST v 1.1) at 6 weeks and 12 weeks, respectively.
Time Frame: 6 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Crizotinib 250 mg BID
Number analyzed (Participants) | 1066
Percentage of participants
  ALK Positive by IUO at Week 6, N=908 | 81.7 [79.0 to 84.2]
  ALK Positive by IUO at Week 12, N=908 | 70.8 [67.7 to 73.8]
  ALK Positive by non-IUO at Week 6, N=158 | 69.6 [61.8 to 76.7]
  ALK Positive by non-IUO at Week 12, N=158 | 61.4 [53.3 to 69.0]

4. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS was defined as the time from the date of the Cycle 1 Day 1 dose to the date of the first documentation of objective tumor progression or death on study due to any cause, whichever occurred first.
Time Frame: 6 years
Population: The safety analysis populations included all participants who received at least 1 dose of study medication (excluding day-7 pharmacokinetic [PK] dosing), and were ALK positive either by IUO (SA-ALK positive by IUO population) or by non-IUO (SA-ALK positive by non-IUO population), respectively.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Crizotinib 250 mg BID
Number analyzed (Participants) | 1066
Months
  ALK Positive by IUO , N= 908 | 8.4 [7.1 to 9.7]
  ALK Positive by non-IUO only , N=158 | 6.9 [5.6 to 9.4]

5. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from the Cycle 1 Day 1 dose to the date of death due to any cause. OS (in months) was calculated as (date of death - date of Cycle 1 Day 1 dose + 1)/30.4.
Time Frame: 6 years
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Crizotinib 250 mg BID
Number analyzed (Participants) | 1066
Months
  ALK-positive by IUO (N= 908) | 21.8 [19.4 to 24.0]
  ALK-positive by non-IUO (N= 158) | 16.9 [13.4 to 21.5]

6. Secondary Outcome: Probability of Survival
Description: Six-month and 1-year survival probabilities were defined as the probabilities of survival at 6 months and 1 year, respectively, after the date of the Cycle 1 Day 1 dose based on the Kaplan-Meier estimate.
Time Frame: 6 years
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of probability
Arm/Group | Crizotinib 250 mg BID
Number analyzed (Participants) | 1066
Percentage of probability
  ALK positive by IUO at 6 Months | 81.7 [79.0 to 84.0]
  ALK positive by non IUO at 6 Months | 77.5 [70.1 to 83.3]
  ALK positive by IUO at 12 Months | 66.5 [63.3 to 69.5]
  ALK positive by non IUO at 12 Months | 62.4 [54.3 to 69.6]

7. Secondary Outcome: Plasma Concentrations of Crizotinib (PF-02341066) and Its Metabolite PF-06260182
Description: Plasma concentrations of crizotinib (PF-02341066) and its metabolite PF-06260182. The method of dispersion is % coefficient of variation.
Time Frame: 6 years
Population: All participants who have ≥ 1 measurement of PF-02341066 or PF-06260182 at the time of reporting are included in PK analysis. Concentration at Cycle 2 Day 1 and beyond are considered steady state, and only included those who received at least 14 continuous days of 250 mg BID dosing.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Crizotinib (PF-02341066): Participants were administered crizotinib at a starting dose of 250 mg orally, BID on a continuous dosing period as two 100-mg tablets and one 50-mg tablet at approximately 12 hours apart the same time each day.
- PF-06260182: PF-06260182 was a PF-02341066 metabolite measured in this study.
Arm/Group | Crizotinib (PF-02341066) | PF-06260182
Number analyzed (Participants) | 906 | 904
ng/mL
  Cycle 1 Day 1 (N= 13, 13) | 1.95 (55) | 0.00601 (167)
  Cycle 2 Day 1 (N=447, 431) | 279 (46) | 76.2 (79)
  Cycle 3 Day 1 (N=398, 385) | 297 (44) | 80.8 (58)
  Cycle 5 Day 1 (N=297, 290) | 294 (48) | 81.4 (61)

8. Secondary Outcome: Molecular Profiling (ALK Status) Descriptive Statistics for ALK Percentage of Positive Cells by Central Laboratory Test (SA [ALK Positive by IUO] Population)
Description: Molecular profiling outcomes included:Types of EML4-ALK fusion variants and ALK protein expression; Although a secondary objective was defined to explore the relationship of ALK gene fusion to the presence of ALK protein and fusion transcript, no additional analyses of ALK fusion variants or ALK protein were performed for technical reasons. Analyses of change from Baseline in the expression of biomarkers relevant to signaling pathways were not performed because paired Baseline and on-treatment (Cycle 2) tumor tissue required for the analysis, which were to be collected on an optional basis, were not available.
Time Frame: 6 years
Population: The safety analysis population included all participants who received at least 1 dose of study medication (excluding day-7 pharmacokinetic [PK] dosing) and were ALK positive by IUO (SA-ALK positive by IUO population)
Measure: Median (Full Range); unit: Percentage of cells
Arm/Group | Crizotinib 250 mg BID
Number analyzed (Participants) | 908
Percentage of cells | 60.0 (21.18) [15.0 to 100.0]

9. Secondary Outcome: Genotypes of Alleles Possibly Associated With Adverse Hepatic Drug Reactions (Pharmacogenomic Evaluable Population)
Description: The frequency of the candidate gene alleles, HLA-DQA1*02:01, HLA-DQB1*02:02, HLA-DRB1*07:01 and TNXB/rs12153855, were measured in alanine transaminase (ALT) Cases and ALT Controls to evaluate if there were statistically significant associations that would support or suggest any predictive (ie, diagnostic) value of these markers in identifying participants who were at increased risk for hepatic toxicity. The frequency of 2 additional HLA gene alleles, HLA-B*57:01 and HLA-DRB1*15:01, were also measured in ALT Cases and ALT Controls. ALT Cases are defined as those patients with a baseline ALT of ≤1xULN and at least one on-treatment ALT assessment of >3x upper limit of normal (ULN), and ALT Controls represent those patients with baseline and on-treatment assessments of ALT of ≤1xULN.
Time Frame: 6 years
Population: The All Genotyped Population was defined as all participants in the safety analysis population who had at least 1 genotype result. The Pharmacogenomic Evaluable (PE) Population was defined as participants in the All Genotyped Population who had an HLA genotype result and were designated as an ALT Case or Control.
Measure: Number; unit: Percentage of participants
Groups:
- Crizotinib 250 mg BID-ALT Cases; Crizotinib 250 mg BID-ALT Controls: Participants were administered crizotinib at a starting dose of 250 milligram [mg] orally, twice daily (BID) on a continuous dosing period as two 100-mg tablets and one 50-mg tablet at approximately 12 hours apart the same time each day.
Arm/Group | Crizotinib 250 mg BID-ALT Cases | Crizotinib 250 mg BID-ALT Controls
Number analyzed (Participants) | 74 | 115
Percentage of participants
  HLA-DQA1*02:01 | 20.3 | 20.0
  HLA-DQB1*02:02 | 17.6 | 16.5
  HLA-DRB1*07:01 | 20.3 | 20.0
  TNXB/rs12153855 | 10.8 | 16.5
  HLA-B*57:01 | 2.7 | 4.3
  HLA-DRB1*15:01 | 17.6 | 20.9

10. Secondary Outcome: QTc Prolongation in Participants
Description: The percentage of participants with maximum post-dose QTcF/QTcB (<450, 450 - <480, 480 - <500, and ≥500 msec) were evaluated.
Time Frame: 6 years
Population: Participants from the SA population who had a Baseline (last ECG [electrocardiogram] prior to Cycle 1 Day 1 dose) and ≥1 post Baseline ECG measurement and were not included in the ECG sub-study.
Measure: Number; unit: Percentage of participants
Arm/Group | Crizotinib 250 mg BID
Number analyzed (Participants) | 999
Percentage of participants
  Maximum QTcF Interval (<450) | 89.8
  Maximum QTcF Interval (450-<480) | 7.7
  Maximum QTcF Interval (480 - <500) | 1.0
  Maximum QTcF Interval (≥500) | 1.5
  Maximum QTcB Interval (<450) | 74.3
  Maximum QTcB Interval (450-<480) | 21.2
  Maximum QTcB Interval (480-<500) | 2.4
  Maximum QTcB Interval (≥500) | 2.1

11. Secondary Outcome: Mean Change From Baseline in QLQ-C30 Global Quality of Life Scores.
Description: The EORTC QLQ-C30 consists of 30 questions which assess five functional domains (physical, role, cognitive, emotional, and social), global health status/quality of life, disease/treatment related symptoms (fatigue, pain, nausea/vomiting, dyspnea, appetite loss, sleep disturbance, constipation, and diarrhoea), and the perceived financial impact of disease. n is the number of participants who completed the scale at baseline and at the respective Cycle. The subscales of the EORTC QLQ-C30 were scored based on the EORTC scoring manual. The transformed scores range from 0-100. Higher scores indicate higher ("worse") symptom severity, higher ("better") functioning, and better global QoL. Negative change from Baseline scores indicate an improvement in symptoms, decreased functioning, or decreased QoL, while positive change scores indicate an increase in functioning, increased QoL, or deterioration in symptoms.
Time Frame: 6 years
Population: The patient reported outcomes (PRO) evaluable population was defined as the participants from the safety analysis (SA) population who completed a baseline assessment and at least one post-baseline assessment.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Crizotinib 250 mg BID
Number analyzed (Participants) | 976
Units on a scale
  CYCLE2/DAY1 (n=929) | 7.9 (22.2)
  CYCLE3/DAY1 (n=872) | 10.6 (23.7)
  CYCLE4/DAY1 (n=828) | 12.2 (24.9)
  CYCLE5/DAY1 (n=806) | 11.5 (23.9)
  CYCLE6/DAY1 (n=774) | 11.9 (24.8)
  CYCLE7/DAY1 (n=734) | 12.3 (24.7)
  CYCLE8/DAY1 (n=699) | 12.3 (24.1)
  CYCLE9/DAY1 (n=665) | 11.8 (23.5)
  CYCLE10/DAY1 (n=631) | 11.5 (23.6)
  CYCLE11/DAY1 (n=570) | 10.4 (23.9)
  CYCLE12/DAY1 (n=411) | 10.1 (21.6)
  CYCLE13/DAY1 (n=512) | 11.0 (24.0)
  CYCLE14/DAY1 (n=353) | 10.4 (21.5)
  CYCLE15/DAY1 (n=462) | 9.5 (23.9)
  CYCLE16/DAY1 (n=294) | 7.4 (23.2)
  CYCLE17/DAY1 (n=419) | 8.0 (24.3)
  CYCLE18/DAY1 (n=247) | 7.8 (22.0)
  CYCLE19/DAY1 (n=376) | 7.8 (23.1)
  CYCLE20/DAY1 (n=222) | 9.1 (22.4)
  CYCLE21/DAY1 (n=340) | 7.8 (22.5)
  CYCLE22/DAY1 (n=179) | 5.9 (23.7)
  CYCLE23/DAY1 (n=305) | 6.7 (24.0)
  CYCLE24/DAY1 (n=154) | 6.4 (25.0)
  CYCLE25/DAY1 (n=293) | 4.7 (23.3)
  CYCLE26/DAY1 (n=127) | 8.3 (24.7)
  CYCLE27/DAY1 (n=269) | 5.9 (23.2)
  CYCLE28/DAY1 (n=120) | 6.7 (24.2)
  CYCLE29/DAY1 (n=247) | 5.7 (23.3)
  CYCLE30/DAY1 (n=105) | 6.4 (24.9)
  End of treatment (n=450) | -1.0 (27.2)

12. Secondary Outcome: Mean Change From Baseline of EORTC QLQ-C30 Functional and Symptom Scale Scores
Description: The EORTC QLQ-C30 consists of 30 questions which assess five functional domains (physical, role, cognitive, emotional, and social), global health status/quality of life, disease/treatment related symptoms (fatigue, pain, nausea/vomiting, dyspnoea, appetite loss, sleep disturbance, constipation, and diarrhoea), and the perceived financial impact of disease. n is the number of participants who completed the scale at baseline and at the respective Cycle. The subscales of the EORTC QLQ-C30 were scored based on the EORTC scoring manual. The transformed scores range from 0-100. Higher scores indicate higher ("worse") symptom severity, higher ("better") functioning, and better global QoL. Negative change from Baseline scores indicate an improvement in symptoms, decreased functioning, or decreased QoL, while positive change scores indicate an increase in functioning, increased QoL, or deterioration in symptoms.
Time Frame: 6 years
Population: The PRO evaluable population was defined as the participants from the SA population who completed a baseline assessment and at least one post-baseline assessment.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Crizotinib 250 mg BID
Number analyzed (Participants) | 976
Units on a scale
  Physical Functioning (Cycle 2/Day 1) (n=936) | 4.3 (17.1)
  Physical Functioning (Cycle 3/Day 1) (n=879) | 6.6 (18.6)
  Physical Functioning (Cycle 4/Day 1) (n=836) | 8.2 (19.1)
  Physical Functioning (Cycle 5/Day 1) (n=810) | 8.8 (18.8)
  Physical Functioning (Cycle 6/Day 1) (n=778) | 9.5 (18.6)
  Physical Functioning (Cycle 7/Day 1) (n=739) | 10.0 (19.3)
  Physical Functioning (Cycle 8/Day 1) (n= 704) | 10.1 (18.8)
  Physical Functioning (Cycle 9/Day 1) (n= 673) | 10.5 (18.2)
  Physical Functioning (Cycle 10/Day 1) (n= 637) | 9.5 (17.9)
  Physical Functioning (Cycle 11/Day 1) (n=577) | 9.1 (17.9)
  Physical Functioning (Cycle 12/Day 1) (n=412) | 8.2 (17.3)
  Physical Functioning (Cycle 13/Day 1) (n=517) | 8.7 (18.1)
  Physical Functioning (Cycle 14/Day 1) (n=358) | 8.2 (16.5)
  Physical Functioning (Cycle 15/Day 1) (n=466) | 7.3 (19.2)
  Physical Functioning (Cycle 16/Day 1) (n=295) | 6.3 (19.1)
  Physical Functioning (Cycle 17/Day 1) (n=424) | 6.0 (18.9)
  Physical Functioning (Cycle 18/Day 1) (n=250) | 6.1 (18.4)
  Physical Functioning (Cycle 19/Day 1) (n=380) | 6.6 (16.8)
  Physical Functioning (Cycle 20/Day 1) (n=224) | 5.1 (16.8)
  Physical Functioning (Cycle 21/Day 1) (n=346) | 5.7 (17.6)
  Physical Functioning (Cycle 22/Day 1) (n=182) | 3.8 (17.0)
  Physical Functioning (Cycle 23/Day 1) (n=311) | 3.7 (17.1)
  Physical Functioning (Cycle 24/Day 1) (n=156) | 2.4 (18.9)
  Physical Functioning (Cycle 25/Day 1) (n=296) | 4.0 (18.0)
  Physical Functioning (Cycle 26/Day 1) (n=129) | 5.3 (18.1)
  Physical Functioning (Cycle 27/Day 1) (n=275) | 3.8 (16.1)
  Physical Functioning (Cycle 28/Day 1) (n=121) | 3.6 (20.4)
  Physical Functioning (Cycle 29/Day 1) (n=251) | 3.7 (15.8)
  Physical Functioning (Cycle 30/Day 1) (n=109) | 2.8 (21.9)
  Physical Functioning (End of treatment) (n=451) | 0.1 (25.0)
  Cognitive functioning (Cycle 2/Day 1) (n=930) | 1.0 (18.4)
  Cognitive Functioning (Cycle 3/Day 1) (n=874) | 2.1 (19.4)
  Cognitive Functioning (Cycle 4/Day 1) (n=829) | 2.1 (18.6)
  Cognitive Functioning (Cycle 5/Day 1) (n=806) | 2.3 (18.4)
  Cognitive Functioning (Cycle 6/Day 1) (n=773) | 2.5 (18.2)
  Cognitive Functioning (Cycle 7/Day 1) (n=734) | 3.2 (18.6)
  Cognitive Functioning (Cycle 8/Day 1) (n=699) | 3.3 (18.5)
  Cognitive Functioning (Cycle 9/Day 1) (n=667) | 3.0 (18.4)
  Cognitive Functioning (Cycle 10/Day 1) (n=632) | 2.7 (19.0)
  Cognitive Functioning (Cycle 11/Day 1) (n=571) | 3.0 (18.5)
  Cognitive Functioning (Cycle 12/Day 1) (n=411) | 1.5 (17.1)
  Cognitive Functioning (Cycle 13/Day 1) (n=512) | 2.0 (19.3)
  Cognitive Functioning (Cycle 14/Day 1) (n=352) | 1.2 (17.8)
  Cognitive Functioning (Cycle 15/Day 1) (n=462) | 1.3 (19.7)
  Cognitive Functioning (Cycle 16/Day 1) (n=294) | -0.1 (18.1)
  Cognitive Functioning (Cycle 17/Day 1) (n=419) | 0.0 (19.4)
  Cognitive Functioning (Cycle 18/Day 1) (n=247) | 0.1 (19.2)
  Cognitive Functioning (Cycle 19/Day 1) (n=376) | 0.1 (19.2)
  Cognitive Functioning (Cycle 20/Day 1) (n=222) | 0.9 (18.1)
  Cognitive Functioning (Cycle 21/Day 1) (n=340) | -0.1 (17.8)
  Cognitive Functioning (Cycle 22/Day 1) (n=179) | -1.1 (17.5)
  Cognitive Functioning (Cycle 23/Day 1) (n=305) | -0.3 (17.6)
  Cognitive Functioning (Cycle 24/Day 1) (n=154) | -3.6 (21.2)
  Cognitive Functioning (Cycle 25/Day 1) (n=293) | -1.3 (18.1)
  Cognitive Functioning (Cycle 26/Day 1) (n=127) | -0.3 (20.2)
  Cognitive Functioning (Cycle 27/Day 1) (n=269) | -0.9 (17.7)
  Cognitive Functioning (Cycle 28/Day 1) (n=120) | -0.6 (20.7)
  Cognitive Functioning (Cycle 29/Day 1) (n=247) | -0.2 (16.0)
  Cognitive Functioning (Cycle 30/Day 1) (n=106) | -2.5 (23.7)
  Cognitive Functioning (End of treatment) (n=449) | -2.3 (21.7)
  Emotional Functioning (Cycle 2/Day 1) (n=928) | 5.5 (18.4)
  Emotional Functioning (Cycle 3/Day 1) (n=873) | 6.8 (18.8)
  Emotional Functioning (Cycle 4/Day 1) (n=827) | 8.2 (18.3)
  Emotional Functioning (Cycle 5/Day 1) (n=804) | 7.8 (18.3)
  Emotional Functioning (Cycle 6/Day 1) (n=772) | 8.6 (18.0)
  Emotional Functioning (Cycle 7/Day 1) (n=731) | 8.3 (18.3)
  Emotional Functioning (Cycle 8/Day 1) (n=697) | 9.2 (18.9)
  Emotional Functioning (Cycle 9/Day 1) (n=665) | 8.7 (18.6)
  Emotional Functioning (Cycle 10/Day 1) (n=630) | 8.5 (18.9)
  Emotional Functioning (Cycle 11/Day 1) (n=571) | 8.5 (17.6)
  Emotional Functioning (Cycle 12/Day 1) (n=410) | 8.4 (17.6)
  Emotional Functioning (Cycle 13/Day 1) (n=511) | 8.5 (19.1)
  Emotional Functioning (Cycle 14/Day 1) (n=352) | 7.9 (16.6)
  Emotional Functioning (Cycle 15/Day 1) (n=461) | 8.3 (18.7)
  Emotional Functioning (Cycle 16/Day 1) (n=293) | 7.5 (16.8)
  Emotional Functioning (Cycle 17/Day 1) (n=418) | 6.9 (19.2)
  Emotional Functioning (Cycle 18/Day 1) (n=246) | 7.5 (17.2)
  Emotional Functioning (Cycle 19/Day 1) (n=376) | 7.4 (18.3)
  Emotional Functioning (Cycle 20/Day 1) (n=221) | 7.4 (17.6)
  Emotional Functioning (Cycle 21/Day 1) (n=340) | 6.7 (17.5)
  Emotional Functioning (Cycle 22/Day 1) (n=178) | 5.2 (17.9)
  Emotional Functioning (Cycle 23/Day 1) (n=305) | 6.6 (17.6)
  Emotional Functioning (Cycle 24/Day 1) (n=153) | 4.4 (19.5)
  Emotional Functioning (Cycle 25/Day 1) (n=293) | 6.2 (17.4)
  Emotional Functioning (Cycle 26/Day 1) (n=126) | 7.5 (18.9)
  Emotional Functioning (Cycle 27/Day 1) (n=269) | 6.3 (17.6)
  Emotional Functioning (Cycle 28/Day 1) (n=119) | 4.1 (19.2)
  Emotional Functioning (Cycle 29/Day 1) (n=247) | 5.9 (17.7)
  Emotional Functioning (Cycle 30/Day 1) (n=105) | 3.2 (21.5)
  Emotional Functioning (End of treatment) (n=448) | 1.9 (22.3)
  Role Functioning (Cycle 2/Day 1) (n=935) | 4.2 (25.0)
  Role Functioning (Cycle 3/Day 1) (n=879) | 7.3 (27.8)
  Role Functioning (Cycle 4/Day 1) (n=835) | 9.3 (28.7)
  Role Functioning (Cycle 5/Day 1) (n=809) | 9.5 (28.4)
  Role Functioning (Cycle 6/Day 1) (n=778) | 10.5 (28.7)
  Role Functioning (Cycle 7/Day 1) (n=738) | 10.4 (30.2)
  Role Functioning (Cycle 8/Day 1) (n=702) | 10.8 (28.5)
  Role Functioning (Cycle 9/Day 1) (n=671) | 10.9 (28.1)
  Role Functioning (Cycle 10/Day 1) (n=635) | 10.8 (28.8)
  Role Functioning (Cycle 11/Day 1) (n=576) | 10.0 (29.0)
  Role Functioning (Cycle 12/Day 1) (n=413) | 8.4 (28.0)
  Role Functioning (Cycle 13/Day 1) (n=516) | 9.0 (28.8)
  Role Functioning (Cycle 14/Day 1) (n=358) | 8.4 (26.5)
  Role Functioning (Cycle 15/Day 1) (n=465) | 8.8 (28.7)
  Role Functioning (Cycle 16/Day 1) (n=296) | 6.0 (28.3)
  Role Functioning (Cycle 17/Day 1) (n=424) | 6.1 (30.4)
  Role Functioning (Cycle 18/Day 1) (n=250) | 5.2 (27.8)
  Role Functioning (Cycle 19/Day 1) (n=380) | 8.0 (27.5)
  Role Functioning (Cycle 20/Day 1) (n=224) | 5.8 (25.1)
  Role Functioning (Cycle 21/Day 1) (n=346) | 5.3 (27.1)
  Role Functioning (Cycle 22/Day 1) (n=182) | 4.1 (26.7)
  Role Functioning (Cycle 23/Day 1) (n=311) | 3.2 (27.9)
  Role Functioning (Cycle 24/Day 1) (n=157) | 2.7 (29.5)
  Role Functioning (Cycle 25/Day 1) (n=297) | 2.2 (27.2)
  Role Functioning (Cycle 26/Day 1) (n=129) | 6.1 (28.0)
  Role Functioning (Cycle 27/Day 1) (n=275) | 2.4 (27.6)
  Role Functioning (Cycle 28/Day 1) (n=121) | 1.5 (30.0)
  Role Functioning (Cycle 29/Day 1)(n=251) | 1.6 (24.6)
  Role Functioning (Cycle 30/Day 1) (n=109) | 1.1 (34.0)
  Role Functioning (End of treatment) (n=451) | -1.6 (31.9)
  Social Functioning (Cycle 2/Day 1) (n=928) | 6.8 (25.9)
  Social Functioning (Cycle 3/Day 1) (n=872) | 9.1 (26.2)
  Social Functioning (Cycle 4/Day 1) (n=828) | 10.4 (27.2)
  Social Functioning (Cycle 5/Day 1) (n=805) | 10.6 (26.7)
  Social Functioning (Cycle 6/Day 1) (n=773) | 11.1 (27.0)
  Social Functioning (Cycle 7/Day 1) (n=733) | 12.1 (26.5)
  Social Functioning (Cycle 8/Day 1) (n=698) | 12.3 (26.4)
  Social Functioning (Cycle 9/Day 1) (n=666) | 12.0 (26.4)
  Social Functioning (Cycle 10/Day 1) (n=631) | 11.8 (26.1)
  Social Functioning (Cycle 11/Day 1) (n=570) | 12.1 (27.3)
  Social Functioning (Cycle 12/Day 1) (n=410) | 10.3 (26.3)
  Social Functioning (Cycle 13/Day 1) (n=512) | 10.6 (27.3)
  Social Functioning (Cycle 14/Day 1) (n=352) | 10.4 (25.1)
  Social Functioning (Cycle 15/Day 1) (n=462) | 10.1 (28.1)
  Social Functioning (Cycle 16/Day 1) (n=293) | 9.0 (26.4)
  Social Functioning (Cycle 17/Day 1) (n=418) | 8.8 (26.9)
  Social Functioning (Cycle 18/Day 1) (n=246) | 6.6 (25.4)
  Social Functioning (Cycle 19/Day 1) (n=376) | 8.0 (25.6)
  Social Functioning (Cycle 20/Day 1) (n=221) | 5.7 (23.9)
  Social Functioning (Cycle 21/Day 1) (n=340) | 6.7 (26.6)
  Social Functioning (Cycle 22/Day 1) (n=178) | 5.3 (22.7)
  Social Functioning (Cycle 23/Day 1) (n=305) | 7.0 (24.9)
  Social Functioning (Cycle 24/Day 1) (n=153) | 3.6 (26.5)
  Social Functioning (Cycle 25/Day 1) (n=293) | 4.4 (25.8)
  Social Functioning (Cycle 26/Day 1) (n=126) | 5.2 (26.6)
  Social Functioning (Cycle 27/Day 1) (n=269) | 5.3 (26.4)
  Social Functioning (Cycle 28/Day 1) (n=119) | 2.1 (31.4)
  Social Functioning (Cycle 29/Day 1) (n=247) | 6.6 (24.1)
  Social Functioning (Cycle 30/Day 1) (n=105) | 1.6 (29.0)
  Social Functioning (End of treatment) (n=449) | 2.7 (31.2)
  Appetite loss (Cycle 2/Day 1) (n=936) | -2.1 (30.3)
  Appetite loss (Cycle 3/Day 1) (n=877) | -6.3 (31.7)
  Appetite loss (Cycle 4/Day 1) (n=833) | -9.1 (31.9)
  Appetite loss (Cycle 5/Day 1) (n=810) | -10.4 (31.9)
  Appetite loss (Cycle 6/Day 1) (n=778) | -11.4 (32.1)
  Appetite loss (Cycle 7/Day 1) (n=738) | -11.4 (32.4)
  Appetite loss (Cycle 8/Day 1) (n=704) | -11.5 (32.6)
  Appetite loss (Cycle 9/Day 1) (n=673) | -11.7 (32.5)
  Appetite loss (Cycle 10/Day 1) (n=637) | -11.9 (30.9)
  Appetite loss (Cycle 11/Day 1) (n=577) | -11.2 (30.4)
  Appetite loss (Cycle 12/Day 1) (n=413) | -9.1 (30.9)
  Appetite loss (Cycle 13/Day 1) (n=517) | -11.3 (29.8)
  Appetite loss (Cycle 14/Day 1) (n=358) | -9.9 (31.8)
  Appetite loss (Cycle 15/Day 1) (n=466) | -10.5 (30.6)
  Appetite loss (Cycle 16/Day 1) (n=296) | -10.4 (32.4)
  Appetite loss (Cycle 17/Day 1) (n=424) | -8.6 (29.5)
  Appetite loss (Cycle 18/Day 1) (n=250) | -10.1 (31.5)
  Appetite loss (Cycle 19/Day 1) (n=380) | -8.9 (30.9)
  Appetite loss (Cycle 20/Day 1) (n=224) | -12.8 (29.0)
  Appetite loss (Cycle 21/Day 1) (n=346) | -7.5 (30.6)
  Appetite loss (Cycle 22/Day 1) (n=181) | -9.2 (27.7)
  Appetite loss (Cycle 23/Day 1) (n=310) | -4.9 (28.5)
  Appetite loss (Cycle 24/Day 1) (n=157) | -10.9 (30.1)
  Appetite loss (Cycle 25/Day 1) (n=297) | -4.6 (29.0)
  Appetite loss (Cycle 26/Day 1) (n=129) | -12.1 (32.3)
  Appetite loss (Cycle 27/Day 1) (n=275) | -4.2 (29.4)
  Appetite loss (Cycle 28/Day 1) (n=121) | -6.6 (34.6)
  Appetite loss (Cycle 29/Day 1) (n=251) | -3.2 (27.0)
  Appetite loss (Cycle 30/Day 1) (n=109) | -7.6 (29.3)
  Appetite loss (End of treatment) (n=451) | -0.0 (36.9)
  Constipation (Cycle 2/Day 1) (n=929) | 15.4 (32.9)
  Constipation (Cycle 3/Day 1) (n=870) | 10.9 (33.8)
  Constipation (Cycle 4/Day 1) (n=827) | 7.0 (31.0)
  Constipation (Cycle 5/Day 1) (n=804) | 5.5 (30.4)
  Constipation (Cycle 6/Day 1) (n=771) | 5.4 (30.3)
  Constipation (Cycle 7/Day 1) (n=732) | 4.7 (30.3)
  Constipation (Cycle 8/Day 1) (n=698) | 4.5 (29.8)
  Constipation (Cycle 9/Day 1) (n=665) | 5.0 (29.9)
  Constipation (Cycle 10/Day 1) (n=631) | 3.8 (30.0)
  Constipation (Cycle 11/Day 1) (n=571) | 5.2 (29.7)
  Constipation (Cycle 12/Day 1) (n=410) | 6.4 (29.6)
  Constipation (Cycle 13/Day 1) (n=513) | 5.2 (29.0)
  Constipation (Cycle 14/Day 1) (n=349) | 5.0 (28.7)
  Constipation (Cycle 15/Day 1) (n=464) | 6.0 (30.1)
  Constipation (Cycle 16/Day 1) (n=291) | 4.4 (29.9)
  Constipation (Cycle 17/Day 1) (n=420) | 8.3 (30.5)
  Constipation (Cycle 18/Day 1) (n=246) | 6.0 (30.7)
  Constipation (Cycle 19/Day 1) (n=376) | 7.4 (30.5)
  Constipation (Cycle 20/Day 1) (n=221) | 5.9 (33.2)
  Constipation (Cycle 21/Day 1) (n=340) | 7.7 (31.3)
  Constipation (Cycle 22/Day 1) (n=178) | 6.2 (31.2)
  Constipation (Cycle 23/Day 1) (n=306) | 9.7 (31.9)
  Constipation (Cycle 24/Day 1) (n=154) | 9.0 (34.2)
  Constipation (Cycle 25/Day 1) (n=293) | 10.9 (29.4)
  Constipation (Cycle 26/Day 1) (n=126) | 5.6 (32.0)
  Constipation (Cycle 27/Day 1) (n=269) | 8.3 (30.7)
  Constipation (Cycle 28/Day 1) (n=119) | 9.8 (31.1)
  Constipation (Cycle 29/Day 1) (n=247) | 7.8 (29.3)
  Constipation (Cycle 30/Day 1) (n=105) | 11.7 (31.3)
  Constipation (End of treatment) (n=444) | 8.9 (33.0)
  Diarrhea (Cycle 2/Day 1) (n=927) | 11.4 (25.9)
  Diarrhea (Cycle 3/Day 1) (n=872) | 12.8 (26.9)
  Diarrhea (Cycle 4/Day 1) (n=826) | 11.7 (25.6)
  Diarrhea (Cycle 5/Day 1) (n=805) | 12.6 (26.1)
  Diarrhea (Cycle 6/Day 1) (n=772) | 11.6 (26.4)
  Diarrhea (Cycle 7/Day 1) (n=732) | 10.9 (26.3)
  Diarrhea (Cycle 8/Day 1) (n=698) | 9.8 (25.6)
  Diarrhea (Cycle 9/Day 1) (n=665) | 10.5 (25.6)
  Diarrhea (Cycle 10/Day 1) (n=632) | 11.1 (26.6)
  Diarrhea (Cycle 11/Day 1) (n=570) | 10.1 (25.9)
  Diarrhea (Cycle 12/Day 1) (n=411) | 8.1 (25.2)
  Diarrhea (Cycle 13/Day 1) (n=512) | 8.8 (24.0)
  Diarrhea (Cycle 14/Day 1) (n=352) | 10.1 (22.4)
  Diarrhea (Cycle 15/Day 1) (n=461) | 8.5 (23.1)
  Diarrhea (Cycle 16/Day 1) (n=293) | 10.0 (22.5)
  Diarrhea (Cycle 17/Day 1) (n=419) | 8.6 (23.9)
  Diarrhea (Cycle 18/Day 1) (n=247) | 7.4 (22.4)
  Diarrhea (Cycle 19/Day 1) (n=376) | 7.8 (22.5)
  Diarrhea (Cycle 20/Day 1) (n=222) | 6.8 (22.6)
  Diarrhea (Cycle 21/Day 1) (n=340) | 6.6 (20.3)
  Diarrhea (Cycle 22/Day 1) (n=179) | 6.8 (24.2)
  Diarrhea (Cycle 23/Day 1) (n=305) | 8.7 (22.7)
  Diarrhea (Cycle 24/Day 1) (n=154) | 6.4 (23.1)
  Diarrhea (Cycle 25/Day 1) (n=293) | 10.1 (23.4)
  Diarrhea (Cycle 26/Day 1) (n=127) | 5.0 (23.8)
  Diarrhea (Cycle 27/Day 1) (n=269) | 8.3 (24.5)
  Diarrhea (Cycle 28/Day 1) (n=119) | 5.6 (20.5)
  Diarrhea (Cycle 29/Day 1) (n=247) | 9.7 (22.6)
  Diarrhea (Cycle 30/Day 1) (n=106) | 10.1 (25.3)
  Diarrhea (End of treatment) (n=449) | 5.9 (24.5)
  Dyspnoea (Cycle 2/Day 1) (n=933) | -9.8 (26.2)
  Dyspnoea (Cycle 3/Day 1) (n=876) | -11.4 (28.2)
  Dyspnoea (Cycle 4/Day 1) (n=834) | -12.3 (28.6)
  Dyspnoea (Cycle 5/Day 1) (n=808) | -12.2 (27.7)
  Dyspnoea (Cycle 6/Day 1) (n=776) | -13.7 (27.6)
  Dyspnoea (Cycle 7/Day 1) (n=737) | -13.8 (27.8)
  Dyspnoea (Cycle 8/Day 1) (n=702) | -13.8 (28.2)
  Dyspnoea (Cycle 9/Day 1) (n=671) | -13.3 (27.9)
  Dyspnoea (Cycle 10/Day 1) (n=635) | -13.4 (27.6)
  Dyspnoea (Cycle 11/Day 1) (n=575) | -15.0 (27.8)
  Dyspnoea (Cycle 12/Day 1) (n=411) | -13.1 (26.8)
  Dyspnoea (Cycle 13/Day 1) (n=515) | -13.1 (28.1)
  Dyspnoea (Cycle 14/Day 1) (n=356) | -12.7 (27.5)
  Dyspnoea (Cycle 15/Day 1) (n=463) | -12.6 (28.5)
  Dyspnoea (Cycle 16/Day 1) (n=295) | -12.2 (27.6)
  Dyspnoea (Cycle 17/Day 1) (n=421) | -11.8 (27.9)
  Dyspnoea (Cycle 18/Day 1) (n=248) | -11.5 (27.4)
  Dyspnoea (Cycle 19/Day 1) (n=377) | -14.2 (28.0)
  Dyspnoea (Cycle 20/Day 1) (n=222) | -9.2 (26.4)
  Dyspnoea (Cycle 21/Day 1) (n=344) | -13.4 (27.1)
  Dyspnoea (Cycle 22/Day 1) (n=181) | -8.8 (26.4)
  Dyspnoea (Cycle 23/Day 1) (n=309) | -10.9 (26.6)
  Dyspnoea (Cycle 24/Day 1) (n=156) | -8.5 (27.3)
  Dyspnoea (Cycle 25/Day 1) (n=295) | -10.5 (26.3)
  Dyspnoea (Cycle 26/Day 1) (n=129) | -10.1 (27.2)
  Dyspnoea (Cycle 27/Day 1) (n=273) | -9.3 (24.8)
  Dyspnoea (Cycle 28/Day 1) (n=121) | -12.1 (28.9)
  Dyspnoea (Cycle 29/Day 1) (n=249) | -8.8 (25.4)
  Dyspnoea (Cycle 30/Day 1) (n=109) | -11.6 (27.7)
  Dyspnoea (End of treatment) (n=450) | -4.2 (32.8)
  Fatigue (Cycle 2/Day 1) (n=936) | -4.8 (21.8)
  Fatigue (Cycle 3/Day 1) (n=879) | -8.9 (23.7)
  Fatigue (Cycle 4/Day 1) (n=836) | -11.4 (24.1)
  Fatigue (Cycle 5/Day 1) (n=810) | -12.0 (24.2)
  Fatigue (Cycle 6/Day 1) (n=778) | -13.7 (24.3)
  Fatigue (Cycle 7/Day 1) (n=739) | -14.0 (24.6)
  Fatigue (Cycle 8/Day 1) (n=704) | -15.3 (23.7)
  Fatigue (Cycle 9/Day 1) (n=671) | -14.9 (24.0)
  Fatigue (Cycle 10/Day 1) (n=637) | -14.4 (24.2)
  Fatigue (Cycle 11/Day 1) (n=577) | -13.7 (24.3)
  Fatigue (Cycle 12/Day 1) (n=413) | -12.2 (23.4)
  Fatigue (Cycle 13/Day 1) (n=517) | -13.4 (23.6)
  Fatigue (Cycle 14/Day 1) (n=358) | -13.2 (22.3)
  Fatigue (Cycle 15/Day 1) (n=466) | -13.1 (23.9)
  Fatigue (Cycle 16/Day 1) (n=296) | -11.3 (24.1)
  Fatigue (Cycle 17/Day 1) (n=424) | -11.3 (24.6)
  Fatigue (Cycle 18/Day 1) (N=250) | -10.4 (25.2)
  Fatigue (Cycle 19/Day 1) (n=380) | -11.9 (23.7)
  Fatigue (Cycle 20/Day 1) (n=224) | -10.6 (23.2)
  Fatigue (Cycle 21/Day 1) (n=346) | -11.0 (25.0)
  Fatigue (Cycle 22/Day 1) (n=182) | -8.4 (23.0)
  Fatigue (Cycle 23/Day 1) (n=311) | -8.7 (23.3)
  Fatigue (Cycle 24/Day 1) (n=157) | -6.7 (24.1)
  Fatigue (Cycle 25/Day 1) (n=297) | -7.9 (23.2)
  Fatigue (Cycle 26/Day 1) (n=129) | -12.1 (24.8)
  Fatigue (Cycle 27/Day 1) (n=275) | -7.0 (22.3)
  Fatigue (Cycle 28/Day 1) (n=121) | -6.7 (25.2)
  Fatigue (Cycle 29/Day 1) (n=251) | -7.1 (22.1)
  Fatigue (Cycle 30/Day 1) (n=109) | -7.2 (27.0)
  Fatigue (End of treatment) (n=451) | -5.3 (27.5)
  Financial Difficulties (Cycle 2/Day 1) (n=928) | -4.6 (24.1)
  Financial Difficulties (Cycle 3/Day 1) (n=871) | -4.2 (25.2)
  Financial Difficulties (Cycle 4/Day 1) (n=827) | -5.9 (25.7)
  Financial Difficulties (Cycle 5/Day 1) (n=803) | -5.1 (25.6)
  Financial Difficulties (Cycle 6/Day 1) (n=772) | -5.5 (25.4)
  Financial Difficulties (Cycle 7/Day 1) (n=732) | -6.2 (25.8)
  Financial Difficulties (Cycle 8/Day 1) (n=697) | -6.4 (26.0)
  Financial Difficulties (Cycle 9/Day 1) (n=663) | -5.8 (25.8)
  Financial Difficulties (Cycle 10/Day 1) (n=631) | -7.4 (25.0)
  Financial Difficulties (Cycle 11/Day 1) (n=569) | -6.6 (25.4)
  Financial Difficulties (Cycle 12/Day 1) (n=410) | -4.8 (25.4)
  Financial Difficulties (Cycle 13/Day 1) (n=512) | -6.3 (25.8)
  Financial Difficulties (Cycle 14/Day 1) (n=352) | -5.8 (25.4)
  Financial Difficulties (Cycle 15/Day 1) (n=461) | -6.1 (26.7)
  Financial Difficulties (Cycle 16/Day 1) (n=294) | -4.0 (23.8)
  Financial Difficulties (Cycle 17/Day 1) (n=418) | -5.5 (26.8)
  Financial Difficulties (Cycle 18/Day 1) (n=247) | -3.8 (25.2)
  Financial Difficulties (Cycle 19/Day 1) (n=376) | -5.9 (26.8)
  Financial Difficulties (Cycle 20/Day 1) (n=220) | -5.2 (25.4)
  Financial Difficulties (Cycle 21/Day 1) (n=339) | -4.2 (25.9)
  Financial Difficulties (Cycle 22/Day 1) (n=177) | -2.1 (23.1)
  Financial Difficulties (Cycle 23/Day 1) (n=304) | -4.4 (24.9)
  Financial Difficulties (Cycle 24/Day 1) (n=153) | -2.8 (27.3)
  Financial Difficulties (Cycle 25/Day 1) (n=292) | -4.6 (24.8)
  Financial Difficulties (Cycle 26/Day 1) (n=126) | -2.9 (26.0)
  Financial Difficulties (Cycle 27/Day 1) (n=268) | -4.8 (25.5)
  Financial Difficulties (Cycle 28/Day 1) (n=119) | -4.2 (29.9)
  Financial Difficulties (Cycle 29/Day 1) (n=247) | -5.5 (25.2)
  Financial Difficulties (Cycle 30/Day 1) (n=105) | -3.5 (26.5)
  Financial Difficulties (End of treatment) (n=447) | -2.2 (27.5)
  Insomnia (Cycle 2/Day 1) (n=934) | -7.6 (29.3)
  Insomnia (Cycle 3/Day 1) (n=878) | -11.3 (30.1)
  Insomnia (Cycle 4/Day 1) (n=833) | -13.0 (29.7)
  Insomnia (Cycle 5/Day 1) (n=808) | -12.8 (29.8)
  Insomnia (Cycle 6/Day 1) (n=778) | -13.3 (31.1)
  Insomnia (Cycle 7/Day 1) (n=739) | -13.9 (29.7)
  Insomnia (Cycle 8/Day 1) (n=703) | -12.6 (29.9)
  Insomnia (Cycle 9/Day 1) (n=673) | -13.2 (28.8)
  Insomnia (Cycle 10/Day 1) (n=637) | -13.2 (29.4)
  Insomnia (Cycle 11/Day 1) (n=576) | -12.2 (30.0)
  Insomnia (Cycle 12/Day 1) (n=413) | -11.3 (29.7)
  Insomnia (Cycle 13/Day 1) (n=516) | -13.0 (29.5)
  Insomnia (Cycle 14/Day 1) (n=358) | -11.7 (30.3)
  Insomnia (Cycle 15/Day 1) (n=464) | -12.4 (30.0)
  Insomnia (Cycle 16/Day 1) (n=296) | -10.9 (31.6)
  Insomnia (Cycle 17/Day 1) (n=424) | -10.8 (29.2)
  Insomnia (Cycle 18/Day 1) (n=250) | -10.4 (30.3)
  Insomnia (Cycle 19/Day 1) (n=379) | -12.6 (28.9)
  Insomnia (Cycle 20/Day 1) (n=224) | -11.5 (27.1)
  Insomnia (Cycle 21/Day 1) (n=346) | -10.2 (27.6)
  Insomnia (Cycle 22/Day 1) (n=182) | -7.9 (25.8)
  Insomnia (Cycle 23/Day 1) (n=311) | -10.5 (27.2)
  Insomnia (Cycle 24/Day 1) (n=157) | -5.7 (28.0)
  Insomnia (Cycle 25/Day 1) (n=296) | -7.7 (28.8)
  Insomnia (Cycle 26/Day 1) (n=129) | -10.9 (29.2)
  Insomnia (Cycle 27/Day 1) (n=274) | -10.1 (27.4)
  Insomnia (Cycle 28/Day 1) (n=121) | -6.9 (32.7)
  Insomnia (Cycle 29/Day 1) (n=251) | -8.4 (28.5)
  Insomnia (Cycle 30/Day 1) (n=109) | -11.3 (32.1)
  Nausea and Vomiting (Cycle 2/Day 1) (n=936) | 6.2 (23.1)
  Nausea and Vomiting (Cycle 3/Day 1) (n=879) | 2.4 (23.3)
  Nausea and Vomiting (Cycle 4/Day 1) (n=836) | 0.3 (22.6)
  Nausea and Vomiting (Cycle 5/Day 1) (n=810) | -0.4 (21.1)
  Nausea and Vomiting (Cycle 6/Day 1) (n=779) | -1.6 (19.9)
  Nausea and Vomiting (Cycle 7/Day 1) (n=739) | -2.3 (21.0)
  Nausea and Vomiting (Cycle 8/Day 1) (n=704) | -1.9 (19.8)
  Nausea and Vomiting (Cycle 9/Day 1) (n=673) | -1.8 (21.2)
  Nausea and Vomiting (Cycle 10/Day 1) (n=637) | -1.4 (21.6)
  Nausea and Vomiting (Cycle 11/Day 1) (n=577) | -1.7 (20.9)
  Nausea and Vomiting (Cycle 12/Day 1) (n=413) | -1.5 (21.8)
  Nausea and Vomiting (Cycle 13/Day 1) (n=517) | -0.7 (21.2)
  Nausea and Vomiting (Cycle 14/Day 1) (n=358) | -0.4 (23.3)
  Nausea and Vomiting (Cycle 15/Day 1) (n=466) | -0.7 (21.2)
  Nausea and Vomiting (Cycle 16/Day 1) (n=296) | -0.8 (19.5)
  Nausea and Vomiting (Cycle 17/Day 1) (n=424) | -0.3 (20.2)
  Nausea and Vomiting (Cycle 18/Day 1) (n=250) | -0.9 (21.7)
  Nausea and Vomiting (Cycle 19/Day 1) (n=380) | -0.3 (20.1)
  Nausea and Vomiting (Cycle 20/Day 1) (n=224) | -2.3 (18.7)
  Nausea and Vomiting (Cycle 21/Day 1) (n=346) | -1.1 (18.6)
  Nausea and Vomiting (Cycle 22/Day 1) (n=182) | 0.2 (19.0)
  Nausea and Vomiting (Cycle 23/Day 1) (n=311) | 0.8 (17.4)
  Nausea and Vomiting (Cycle 24/Day 1) (n=157) | -1.3 (17.4)
  Nausea and Vomiting (Cycle 25/Day 1) (n=297) | 0.6 (18.0)
  Nausea and Vomiting (Cycle 26/Day 1) (n=129) | -2.3 (20.2)
  Nausea and Vomiting (Cycle 27/Day 1) (n=275) | 1.9 (17.5)
  Nausea and Vomiting (Cycle 28/Day 1) (n=121) | 1.8 (19.7)
  Nausea and Vomiting (Cycle 29/Day 1) (n=251) | 2.5 (18.9)
  Nausea and Vomiting (Cycle 30/Day 1) (n=109) | -0.5 (17.5)
  Nausea and Vomiting (End of treatment) (n=451) | 4.0 (25.3)
  Pain (Cycle 2/Day 1) (n=935) | -13.1 (26.6)
  Pain (Cycle 3/Day 1) (n=880) | -16.0 (28.0)
  Pain (Cycle 4/Day 1) (n=836) | -15.7 (27.8)
  Pain (Cycle 5/Day 1) (n=810) | -15.5 (27.4)
  Pain (Cycle 6/Day 1) (n=779) | -15.5 (27.8)
  Pain (Cycle 7/Day 1) (n=739) | -16.0 (29.0)
  Pain (Cycle 8/Day 1) (n=705) | -15.9 (28.5)
  Pain (Cycle 9/Day 1) (n=673) | -15.5 (28.7)
  Pain (Cycle 10/Day 1) (n=637) | -15.1 (27.6)
  Pain (Cycle 11/Day 1) (n=577) | -14.6 (27.6)
  Pain (Cycle 12/Day 1) (n=414) | -13.6 (29.2)
  Pain (Cycle 13/Day 1) (n=517) | -13.8 (28.0)
  Pain (Cycle 14/Day 1) (n=357) | -13.9 (29.5)
  Pain (Cycle 15/Day 1) (n=466) | -12.1 (27.0)
  Pain (Cycle 16/Day 1) (n=296) | -12.5 (27.9)
  Pain (Cycle 17/Day 1) (n=424) | -10.6 (25.6)
  Pain (Cycle 18/Day 1) (n=250) | -11.1 (27.5)
  Pain (Cycle 19/Day 1) (n=380) | -10.8 (24.1)
  Pain (Cycle 20/Day 1) (n=224) | -11.0 (27.2)
  Pain (Cycle 21/Day 1) (n=346) | -10.1 (25.2)
  Pain (Cycle 22/Day 1) (n=182) | -7.7 (26.2)
  Pain (Cycle 23/Day 1) (n=311) | -7.4 (26.0)
  Pain (Cycle 24/Day 1) (n=157) | -8.8 (27.7)
  Pain (Cycle 25/Day 1) (n=297) | -8.8 (24.6)
  Pain (Cycle 26/Day 1) (n=129) | -12.5 (29.5)
  Pain (Cycle 27/Day 1) (n=275) | -7.6 (25.3)
  Pain (Cycle 28/Day 1) (n=121) | -7.9 (32.4)
  Pain (Cycle 29/Day 1) (n=251) | -8.1 (24.6)
  Pain (Cycle 30/Day 1) (n=109) | -7.5 (29.8)
  Pain (End of treatment) (n=451) | -5.3 (31.2)
  Insomnia (End of treatment) 9n=451) | -5.7 (33.6)

13. Secondary Outcome: Mean Change From Baseline of QLQ-LC13 Scale Scores
Description: The QLQ-LC13 consists of 1 multi-item scale and 9 single items that assess specific symptoms (dyspnoea, cough, hemoptysis, and site-specific pain), side effects (sore mouth, dysphagia, neuropathy, and alopecia), and pain medication use of lung cancer patients. n is the number of participants who completed the scale at baseline and at the respective Cycle. The subscales of the EORTC QLQ-LC13 were scored based on the EORTC scoring manual. The transformed scores range from 0-100. Higher scores indicate higher ("worse") symptom severity, higher ("better") functioning, and better global QoL. Negative change from Baseline scores indicate an improvement in symptoms, decreased functioning, or decreased QoL, while positive change scores indicate an increase in functioning, increased QoL, or deterioration in symptoms.
Time Frame: 6 years
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Crizotinib 250 mg BID
Number analyzed (Participants) | 976
Units on a scale
  Alopecia (Cycle 2/Day 1) (n=920) | -9.1 (29.6)
  Alopecia (Cycle 3/Day 1) (n=870) | -10.2 (31.6)
  Alopecia (Cycle 4/Day 1) (n=829) | -11.6 (30.7)
  Alopecia (Cycle 5/Day 1) (n=805) | -12.2 (32.3)
  Alopecia (Cycle 6/Day 1) (n=770) | -10.5 (30.9)
  Alopecia (Cycle 7/Day 1) (n=734) | -11.9 (32.3)
  Alopecia (Cycle 8/Day 1) (n=700) | -11.9 (33.2)
  Alopecia (Cycle 9/Day 1) (n=667) | -11.3 (34.7)
  Alopecia (Cycle 10/Day 1) (n=633) | -10.8 (33.9)
  Alopecia (Cycle 11/Day 1) (n=574) | -11.3 (34.8)
  Alopecia (Cycle 12/Day 1) (n=409) | -7.8 (34.8)
  Alopecia (Cycle 13/Day 1) (n=512) | -10.8 (35.0)
  Alopecia (Cycle 14/Day 1) (n=353) | -8.2 (36.4)
  Alopecia (Cycle 15/Day 1) (n=462) | -11.8 (34.3)
  Alopecia (Cycle 16/Day 1) (n=293) | -7.7 (34.1)
  Alopecia (Cycle 17/Day 1) (n=419) | -9.5 (32.9)
  Alopecia (Cycle 18/Day 1) (n=247) | -6.4 (31.3)
  Alopecia (Cycle 19/Day 1) (n=377) | -8.9 (34.1)
  Alopecia (Cycle 20/Day 1) (n=222) | -9.0 (30.7)
  Alopecia (Cycle 21/Day 1) (n=342) | -7.8 (32.9)
  Alopecia (Cycle 22/Day 1) (n=180) | -7.6 (35.6)
  Alopecia (Cycle 23/Day 1) (n=310) | -7.0 (33.2)
  Alopecia (Cycle 24/Day 1) (n=156) | -4.1 (34.1)
  Alopecia (Cycle 25/Day 1) (n=293) | -8.2 (31.8)
  Alopecia (Cycle 26/Day 1) (n=126) | -4.5 (31.1)
  Alopecia (Cycle 27/Day 1) (n=271) | -8.5 (31.5)
  Alopecia (Cycle 28/Day 1) (n=119) | -3.9 (33.1)
  Alopecia (Cycle 29/Day 1) (n=247) | -9.2 (28.3)
  Alopecia (Cycle 30/Day 1) (n=107) | -5.0 (31.7)
  Alopecia (End of treatment) (n=447) | -9.9 (35.3)
  Coughing (Cycle 2/Day 1) (n=926) | -12.9 (28.8)
  Coughing (Cycle 3/Day 1) (n=879) | -15.5 (31.8)
  Coughing (Cycle 4/Day 1) (n=832) | -17.7 (31.1)
  Coughing (Cycle 5/Day 1) (n=807) | -17.3 (31.8)
  Coughing (Cycle 6/Day 1) (n=775) | -18.3 (32.1)
  Coughing (Cycle 7/Day 1) (n=735) | -20.1 (32.2)
  Coughing (Cycle 8/Day 1) (n=703) | -20.8 (31.8)
  Coughing (Cycle 9/Day 1) (n=669) | -20.2 (30.9)
  Coughing (Cycle 10/Day 1) (n=636) | -19.9 (32.0)
  Coughing (Cycle 11/Day 1) (n=575) | -19.9 (31.6)
  Coughing (Cycle 12/Day 1) (n=414) | -19.2 (29.5)
  Coughing (Cycle 13/Day 1) (n=513) | -18.6 (32.6)
  Coughing (Cycle 14/Day 1) (n=355) | -17.9 (32.1)
  Coughing (Cycle 15/Day 1) (n=461) | -17.8 (31.7)
  Coughing (Cycle 16/Day 1) (n=294) | -17.3 (29.5)
  Coughing (Cycle 17/Day 1) (n=421) | -18.4 (32.5)
  Coughing (Cycle 18/Day 1) (n=249) | -16.9 (33.1)
  Coughing (Cycle 19/Day 1) (n=379) | -18.8 (30.3)
  Coughing (Cycle 20/Day 1) (n=222) | -18.3 (32.7)
  Coughing (Cycle 21/Day 1) (n=343) | -18.0 (31.0)
  Coughing (Cycle 22/Day 1) (n=181) | -16.7 (33.1)
  Coughing (Cycle 23/Day 1) (n=311) | -18.4 (32.1)
  Coughing (Cycle 24/Day 1) (n=155) | -18.9 (31.3)
  Coughing (Cycle 25/Day 1) (n=294) | -18.1 (31.3)
  Coughing (Cycle 26/Day 1) (n=125) | -21.9 (30.8)
  Coughing (Cycle 27/Day 1) (n=272) | -17.8 (32.2)
  Coughing (Cycle 28/Day 1) (n=119) | -19.6 (30.8)
  Coughing (Cycle 29/Day 1) (n=249) | -17.1 (31.3)
  Coughing (Cycle 30/Day 1) (n=106) | -16.7 (29.5)
  Coughing (End of treatment) (n=452) | -11.1 (33.5)
  Dysphagia (Cycle 2/Day 1) (n=926) | 0.0 (19.6)
  Dysphagia (Cycle 3/Day 1) (n=879) | -1.1 (20.1)
  Dysphagia (Cycle 4/Day 1) (n=831) | -2.2 (20.8)
  Dysphagia (Cycle 5/Day 1) (n=807) | -2.3 (20.0)
  Dysphagia (Cycle 6/Day 1) (n=776) | -3.0 (19.9)
  Dysphagia (Cycle 7/Day 1) (n=737) | -3.1 (20.7)
  Dysphagia (Cycle 8/Day 1) (n=702) | -3.1 (18.6)
  Dysphagia (Cycle 9/Day 1) (n=670) | -2.7 (20.2)
  Dysphagia (Cycle 10/Day 1) (n=637) | -2.9 (19.4)
  Dysphagia (Cycle 11/Day 1) (n=577) | -3.0 (19.2)
  Dysphagia (Cycle 12/Day 1) (n=414) | -2.7 (18.1)
  Dysphagia (Cycle 13/Day 1) (n=513) | -3.1 (17.8)
  Dysphagia (Cycle 14/Day 1) (n=355) | -1.7 (18.2)
  Dysphagia (Cycle 15/Day 1) (n=463) | -2.8 (17.5)
  Dysphagia (Cycle 16/Day 1) (n=294) | -1.3 (20.1)
  Dysphagia (Cycle 17/Day 1) (n=422) | -2.2 (19.0)
  Dysphagia (Cycle 18/Day 1) (n=249) | -2.5 (18.4)
  Dysphagia (Cycle 19/Day 1) (n=378) | -2.0 (17.3)
  Dysphagia (Cycle 20/Day 1) (n=223) | -3.4 (18.5)
  Dysphagia (Cycle 21/Day 1) (n=344) | -2.5 (18.2)
  Dysphagia (Cycle 22/Day 1) (n=182) | -1.8 (19.7)
  Dysphagia (Cycle 23/Day 1) (n=311) | -3.4 (17.0)
  Dysphagia (Cycle 24/Day 1) (n=156) | -1.4 (16.5)
  Dysphagia (Cycle 25/Day 1) (n=295) | -2.8 (17.3)
  Dysphagia (Cycle 26/Day 1) (n=126) | -1.1 (15.7)
  Dysphagia (Cycle 27/Day 1) (n=274) | -1.6 (17.5)
  Dysphagia (Cycle 28/Day 1) (n=120) | -1.4 (16.4)
  Dysphagia (Cycle 29/Day 1) (n=248) | -1.5 (16.5)
  Dysphagia (Cycle 30/Day 1) (n=107) | -0.9 (18.0)
  Dysphagia (End of treatment) (n=449) | 1.9 (23.5)
  Dyspnoea (Cycle 2/Day 1) (n=928) | -8.0 (19.0)
  Dyspnoea (Cycle 3/Day 1) (n=878) | -9.7 (21.5)
  Dyspnoea (Cycle 4/Day 1) (n=833) | -10.7 (21.7)
  Dyspnoea (Cycle 5/Day 1) (n=809) | -10.6 (21.4)
  Dyspnoea (Cycle 6/Day 1) (n=775) | -10.6 (21.7)
  Dyspnoea (Cycle 7/Day 1) (n=737) | -11.1 (21.1)
  Dyspnoea (Cycle 8/Day 1) (n=704) | -12.0 (20.7)
  Dyspnoea (Cycle 9/Day 1) (n=669) | -11.0 (20.7)
  Dyspnoea (Cycle 10/Day 1) (n=637) | -10.7 (21.1)
  Dyspnoea (Cycle 12/Day 1) (n=414) | -9.0 (20.2)
  Dyspnoea (Cycle 13/Day 1) (n=514) | -9.8 (21.1)
  Dyspnoea (Cycle 14/Day 1) (n=354) | -9.2 (20.0)
  Dyspnoea (Cycle 15/Day 1) (n=463) | -8.9 (21.6)
  Dyspnoea (Cycle 16/Day 1) (n=293) | -7.7 (21.3)
  Dyspnoea (Cycle 17/Day 1) (n=421) | -7.3 (20.5)
  Dyspnoea (Cycle 18/Day 1) (n=249) | -6.9 (21.3)
  Dyspnoea (Cycle 19/Day 1) (n=379) | -8.6 (19.7)
  Dyspnoea (Cycle 20/Day 1) (n=223) | -5.8 (19.8)
  Dyspnoea (Cycle 21/Day 1) (n=344) | -7.8 (19.5)
  Dyspnoea (Cycle 22/Day 1) (n=182) | -5.6 (18.3)
  Dyspnoea (Cycle 23/Day 1) (n=311) | -6.1 (19.3)
  Dyspnoea (Cycle 24/Day 1) (n=156) | -6.2 (18.3)
  Dyspnoea (Cycle 25/Day 1) (n=295) | -6.1 (19.7)
  Dyspnoea (Cycle 26/Day 1) (n=126) | -6.6 (19.3)
  Dyspnoea (Cycle 27/Day 1) (n=273) | -5.7 (19.0)
  Dyspnoea (Cycle 28/Day 1) (n=120) | -5.8 (19.5)
  Dyspnoea (Cycle 29/Day 1) (n=249) | -3.9 (19.2)
  Dyspnoea (Cycle 30/Day 1) (n=107) | -4.6 (17.5)
  Dyspnoea (End of treatment) (n=448) | -3.0 (25.7)
  Haemoptysis (Cycle 2/Day 1) (n=925) | -2.6 (12.6)
  Haemoptysis (Cycle 3/Day 1) (n=879) | -3.0 (12.6)
  Haemoptysis (Cycle 4/Day 1) (n=833) | -2.9 (12.7)
  Haemoptysis (Cycle 5/Day 1) (n=808) | -2.6 (12.9)
  Haemoptysis (Cycle 6/Day 1) (n=774) | -2.8 (12.0)
  Haemoptysis (Cycle 7/Day 1) (n=735) | -2.9 (12.7)
  Haemoptysis (Cycle 8/Day 1) (n=703) | -3.1 (11.9)
  Haemoptysis (Cycle 9/Day 1) (n=669) | -3.0 (11.7)
  Haemoptysis (Cycle 10/Day 1) (n=635) | -2.6 (11.7)
  Haemoptysis (Cycle 11/Day 1) (n=576) | -2.7 (11.6)
  Haemoptysis (Cycle 12/Day 1) (n=413) | -2.6 (10.3)
  Haemoptysis (Cycle 13/Day 1) (n=514) | -2.1 (12.0)
  Haemoptysis (Cycle 14/Day 1) (n=354) | -2.7 (11.3)
  Haemoptysis (Cycle 15/Day 1) (n=462) | -2.2 (10.8)
  Haemoptysis (Cycle 16/Day 1) (n=294) | -2.5 (11.4)
  Haemoptysis (Cycle 17/Day 1) (n=420) | -1.9 (11.4)
  Haemoptysis (Cycle 18/Day 1) (n=249) | -2.4 (12.1)
  Haemoptysis (Cycle 19/Day 1) (n=378) | -2.1 (11.5)
  Haemoptysis (Cycle 20/Day 1) (n=223) | -2.4 (13.6)
  Haemoptysis (Cycle 21/Day 1) (n=342) | -2.5 (11.5)
  Haemoptysis (Cycle 22/Day 1) (n=182) | -2.9 (11.2)
  Haemoptysis (Cycle 23/Day 1) (n=309) | -2.7 (12.5)
  Haemoptysis (Cycle 24/Day 1) (n=156) | -2.4 (12.0)
  Haemoptysis (Cycle 25/Day 1) (n=294) | -2.8 (12.4)
  Haemoptysis (Cycle 26/Day 1) (n=126) | -3.2 (12.9)
  Haemoptysis (Cycle 27/Day 1) (n=272) | -2.9 (11.4)
  Haemoptysis (Cycle 28/Day 1) (n=119) | -3.1 (12.3)
  Haemoptysis (Cycle 29/Day 1) (n=248) | -1.7 (12.1)
  Haemoptysis (Cycle 30/Day 1) (n=107) | -2.8 (11.3)
  Haemoptysis (End of treatment) (n=451) | -1.4 (15.9)
  Pain in Arm or Shoulder (Cycle 2/Day 1) (n=926) | -9.6 (26.9)
  Pain in Arm or Shoulder (Cycle 3/Day 1) (n=876) | -12.2 (27.0)
  Pain in Arm or Shoulder (Cycle 4/Day 1) (n=832) | -12.5 (28.2)
  Pain in Arm or Shoulder (Cycle 5/Day 1) (n=807) | -11.7 (27.1)
  Pain in Arm or Shoulder (Cycle 6/Day 1) (n=773) | -11.6 (26.3)
  Pain in Arm or Shoulder (Cycle 7/Day 1) (n=738) | -11.3 (28.1)
  Pain in Arm or Shoulder (Cycle 8/Day 1) (n=702) | -11.7 (28.5)
  Pain in Arm or Shoulder (Cycle 9/Day 1) (n=669) | -11.9 (28.5)
  Pain in Arm or Shoulder (Cycle 10/Day 1) (n=635) | -11.3 (28.0)
  Pain in Arm or Shoulder (Cycle 11/Day 1) (n=576) | -12.1 (27.3)
  Pain in Arm or Shoulder (Cycle 12/Day 1) (n=414) | -11.0 (27.7)
  Pain in Arm or Shoulder (Cycle 13/Day 1) (n=513) | -10.9 (27.2)
  Pain in Arm or Shoulder (Cycle 14/Day 1) (n=355) | -11.3 (27.3)
  Pain in Arm or Shoulder (Cycle 15/Day 1) (n=461) | -10.3 (25.6)
  Pain in Arm or Shoulder (Cycle 16/Day 1) (n=293) | -9.9 (28.0)
  Pain in Arm or Shoulder (Cycle 17/Day 1) (n=421) | -8.2 (26.5)
  Pain in Arm or Shoulder (Cycle 18/Day 1) (n=249) | -9.4 (27.6)
  Pain in Arm or Shoulder (Cycle 19/Day 1) (n=379) | -9.1 (26.5)
  Pain in Arm or Shoulder (Cycle 20/Day 1) (n=222) | -7.4 (27.3)
  Pain in Arm or Shoulder (Cycle 21/Day 1) (n=344) | -9.0 (27.0)
  Pain in Arm or Shoulder (Cycle 22/Day 1) (n=182) | -9.0 (29.1)
  Pain in Arm or Shoulder (Cycle 23/Day 1) (n=311) | -8.9 (25.5)
  Pain in Arm or Shoulder (Cycle 24/Day 1) (n=155) | -9.7 (30.6)
  Pain in Arm or Shoulder (Cycle 25/Day 1) (n=295) | -9.2 (26.0)
  Pain in Arm or Shoulder (Cycle 26/Day 1) (n=126) | -10.8 (33.7)
  Pain in Arm or Shoulder (Cycle 27/Day 1) (n=274) | -8.6 (26.5)
  Pain in Arm or Shoulder (Cycle 28/Day 1) (n=119) | -8.7 (29.6)
  Pain in Arm or Shoulder (Cycle 29/Day 1) (n=248) | -7.9 (27.2)
  Pain in Arm or Shoulder (Cycle 30/Day 1) (n=107) | -8.1 (30.3)
  Pain in Arm or Shoulder (End of treatment) (n=445) | -5.8 (30.7)
  Pain in Chest (Cycle 2/Day 1) (n=928) | -9.5 (23.4)
  Pain in Chest (Cycle 3/Day 1) (n=875) | -11.9 (25.1)
  Pain in Chest (Cycle 4/Day 1) (n=833) | -12.1 (26.1)
  Pain in Chest (Cycle 5/Day 1) (n=808) | -11.8 (25.8)
  Pain in Chest (Cycle 6/Day 1) (n=774) | -12.1 (25.3)
  Pain in Chest (Cycle 7/Day 1) (n=735) | -12.6 (25.4)
  Pain in Chest (Cycle 8/Day 1) (n=703) | -13.2 (25.0)
  Pain in Chest (Cycle 9/Day 1) (n=665) | -13.1 (25.8)
  Pain in Chest (Cycle 10/Day 1) (n=633) | -12.9 (26.0)
  Pain in Chest (Cycle 11/Day 1) (n=574) | -12.0 (25.5)
  Pain in Chest (Cycle 12/Day 1) (n=414) | -10.7 (25.5)
  Pain in Chest (Cycle 13/Day 1) (n=513) | -12.6 (24.5)
  Pain in Chest (Cycle 14/Day 1) (n=355) | -11.5 (24.4)
  Pain in Chest (Cycle 15/Day 1) (n=462) | -11.9 (24.7)
  Pain in Chest (Cycle 16/Day 1) (n=294) | -11.0 (23.4)
  Pain in Chest (Cycle 17/Day 1) (n=421) | -11.6 (23.8)
  Pain in Chest (Cycle 18/Day 1) (n=249) | -8.0 (23.1)
  Pain in Chest (Cycle 19/Day 1) (n=378) | -11.2 (23.8)
  Pain in Chest (Cycle 20/Day 1) (n=222) | -9.4 (24.3)
  Pain in Chest (Cycle 21/Day 1) (n=343) | -11.9 (23.5)
  Pain in Chest (Cycle 22/Day 1) (n=182) | -10.1 (21.9)
  Pain in Chest (Cycle 23/Day 1) (n=308) | -10.8 (24.0)
  Pain in Chest (Cycle 24/Day 1) (n=156) | -7.1 (26.8)
  Pain in Chest (Cycle 25/Day 1) (n=293) | -10.2 (22.3)
  Pain in Chest (Cycle 26/Day 1) (n=126) | -10.6 (25.2)
  Pain in Chest (Cycle 27/Day 1) (n=272) | -9.2 (22.0)
  Pain in Chest (Cycle 28/Day 1) (n=120) | -9.4 (26.7)
  Pain in Chest (Cycle 29/Day 1) (n=248) | -9.5 (24.4)
  Pain in Chest (Cycle 30/Day 1) (n=107) | -5.3 (26.8)
  Pain in Chest (End of treatment) (n=451) | -6.7 (28.0)
  Pain in Other Parts (Cycle 2/Day 1) (n=893) | -10.0 (31.3)
  Pain in Other Parts (Cycle 3/Day 1) (n=854) | -12.0 (31.9)
  Pain in Other Parts (Cycle 4/Day 1) (n=806) | -13.5 (31.0)
  Pain in Other Parts (Cycle 5/Day 1) (n=793) | -12.2 (30.2)
  Pain in Other Parts (Cycle 6/Day 1) (n=752) | -12.5 (30.9)
  Pain in Other Parts (Cycle 7/Day 1) (n=715) | -11.8 (30.3)
  Pain in Other Parts (Cycle 8/Day 1) (n=680) | -11.7 (30.5)
  Pain in Other Parts (Cycle 9/Day 1) (n=650) | -13.1 (29.9)
  Pain in Other Parts (Cycle 10/Day 1) (n=616) | -12.1 (30.4)
  Pain in Other Parts (Cycle 11/Day 1) (n=562) | -10.8 (29.3)
  Pain in Other Parts (Cycle 12/Day 1) (n=399) | -11.6 (30.9)
  Pain in Other Parts (Cycle 13/Day 1) (n=499) | -9.9 (30.0)
  Pain in Other Parts (Cycle 14/Day 1) (n=342) | -11.5 (31.3)
  Pain in Other Parts (Cycle 15/Day 1) (n=451) | -10.1 (28.9)
  Pain in Other Parts (Cycle 16/Day 1) (n=282) | -9.6 (30.3)
  Pain in Other Parts (Cycle 17/Day 1) (n=411) | -8.8 (28.1)
  Pain in Other Parts (Cycle 18/Day 1) (n=239) | -8.6 (31.0)
  Pain in Other Parts (Cycle 19/Day 1) (n=370) | -8.8 (29.0)
  Pain in Other Parts (Cycle 20/Day 1) (n=210) | -9.4 (31.3)
  Pain in Other Parts (Cycle 21/Day 1) (n=337) | -8.2 (28.6)
  Pain in Other Parts (Cycle 22/Day 1) (n=176) | -10.4 (30.2)
  Pain in Other Parts (Cycle 23/Day 1) (n=300) | -6.6 (29.2)
  Pain in Other Parts (Cycle 24/Day 1) (n=149) | -7.8 (35.2)
  Pain in Other Parts (Cycle 25/Day 1) (n=286) | -7.2 (30.2)
  Pain in Other Parts (Cycle 26/Day 1) (n=121) | -8.8 (34.6)
  Pain in Other Parts (Cycle 27/Day 1) (n=267) | -5.9 (29.5)
  Pain in Other Parts (Cycle 28/Day 1) (n=116) | -3.2 (34.6)
  Pain in Other Parts (Cycle 29/Day 1) (n=242) | -6.3 (27.1)
  Pain in Other Parts (Cycle 30/Day 1) (n=102) | -6.5 (34.8)
  Pain in Other Parts (End of treatment) (n=427) | -4.6 (34.8)
  Peripheral Neuropathy (Cycle 2/Day 1) (n=925) | 0.6 (25.3)
  Peripheral Neuropathy (Cycle 3/Day 1) (n=876) | -0.4 (25.6)
  Peripheral Neuropathy (Cycle 4/Day 1) (n=833) | -1.7 (26.5)
  Peripheral Neuropathy (Cycle 5/Day 1) (n=807) | -1.2 (26.3)
  Peripheral Neuropathy (Cycle 6/Day 1) (n=775) | -1.4 (26.5)
  Peripheral Neuropathy (Cycle 7/Day 1) (n=737) | -2.6 (27.2)
  Peripheral Neuropathy (Cycle 8/Day 1) (n=703) | -2.1 (25.6)
  Peripheral Neuropathy (Cycle 9/Day 1) (n=668) | -1.8 (27.2)
  Peripheral Neuropathy (Cycle 10/Day 1) (n=635) | -1.0 (26.4)
  Peripheral Neuropathy (Cycle 11/Day 1) (n=575) | -1.6 (27.5)
  Peripheral Neuropathy (Cycle 12/Day 1) (n=413) | -0.8 (27.3)
  Peripheral Neuropathy (Cycle 13/Day 1) (n=512) | -1.5 (27.0)
  Peripheral Neuropathy (Cycle 14/Day 1) (n=354) | -2.1 (28.6)
  Peripheral Neuropathy (Cycle 15/Day 1) (n=462) | -0.7 (27.5)
  Peripheral Neuropathy (Cycle 16/Day 1) (n=294) | -1.5 (29.9)
  Peripheral Neuropathy (Cycle 17/Day 1) (n=418) | -0.3 (28.3)
  Peripheral Neuropathy (Cycle 18/Day 1) (n=249) | -0.7 (28.3)
  Peripheral Neuropathy (Cycle 19/Day 1) (n=378) | -1.5 (23.9)
  Peripheral Neuropathy (Cycle 20/Day 1) (n=221) | -0.0 (28.1)
  Peripheral Neuropathy (Cycle 21/Day 1) (n=342) | 0.2 (27.6)
  Peripheral Neuropathy (Cycle 22/Day 1) (n=182) | -3.7 (27.6)
  Peripheral Neuropathy (Cycle 23/Day 1) (n=310) | -1.0 (26.2)
  Peripheral Neuropathy (Cycle 24/Day 1) (n=156) | -1.7 (26.4)
  Peripheral Neuropathy (Cycle 25/Day 1) (n=295) | 2.3 (25.5)
  Peripheral Neuropathy (Cycle 26/Day 1) (n=126) | -1.6 (24.9)
  Peripheral Neuropathy (Cycle 27/Day 1) (n=274) | 2.1 (27.1)
  Peripheral Neuropathy (Cycle 28/Day 1) (n=119) | -0.6 (27.1)
  Peripheral Neuropathy (Cycle 29/Day 1) (n=249) | 1.5 (26.3)
  Peripheral Neuropathy (Cycle 30/Day 1) (n=107) | -0.6 (28.2)
  Peripheral Neuropathy (End of treatment) (n=451) | -0.6 (26.6)
  Sore Mouth (Cycle 2/Day 1) (n=928) | 1.0 (20.0)
  Sore Mouth (Cycle 3/Day 1) (n=879) | -0.2 (19.8)
  Sore Mouth (Cycle 4/Day 1) (n=834) | -0.6 (19.1)
  Sore Mouth (Cycle 5/Day 1) (n=808) | -1.3 (17.9)
  Sore Mouth (Cycle 6/Day 1) (n=776) | -1.8 (17.1)
  Sore Mouth (Cycle 7/Day 1) (n=738) | -1.2 (18.3)
  Sore Mouth (Cycle 8/Day 1) (n=704) | -2.2 (17.0)
  Sore Mouth (Cycle 9/Day 1) (n=669) | -2.1 (18.3)
  Sore Mouth (Cycle 10/Day 1) (n=636) | -1.7 (19.1)
  Sore Mouth (Cycle 11/Day 1) (n=577) | -1.8 (17.2)
  Sore Mouth (Cycle 12/Day 1) (n=414) | -1.9 (17.1)
  Sore Mouth (Cycle 13/Day 1) (n=514) | -1.5 (18.0)
  Sore Mouth (Cycle 14/Day 1) (n=354) | -1.3 (14.8)
  Sore Mouth (Cycle 15/Day 1) (n=463) | -0.9 (16.1)
  Sore Mouth (Cycle 16/Day 1) (n=294) | 0.1 (16.6)
  Sore Mouth (Cycle 17/Day 1) (n=422) | -1.4 (17.6)
  Sore Mouth (Cycle 18/Day 1) (n=249) | -0.9 (18.0)
  Sore Mouth (Cycle 19/Day 1) (n=379) | -0.9 (17.3)
  Sore Mouth (Cycle 20/Day 1) (n=223) | -1.3 (17.7)
  Sore Mouth (Cycle 21/Day 1) (n=344) | -0.6 (18.0)
  Sore Mouth (Cycle 22/Day 1) (n=182) | -1.1 (14.8)
  Sore Mouth (Cycle 23/Day 1) (n=311) | 0.3 (17.7)
  Sore Mouth (Cycle 24/Day 1) (n=156) | 2.6 (17.2)
  Sore Mouth (Cycle 25/Day 1) (n=294) | -1.6 (17.6)
  Sore Mouth (Cycle 26/Day 1) (n=126) | -2.4 (14.7)
  Sore Mouth (Cycle 27/Day 1) (n=274) | -0.6 (18.4)
  Sore Mouth (Cycle 28/Day 1) (n=120) | -0.3 (15.3)
  Sore Mouth (Cycle 29/Day 1) (n=249) | -1.7 (16.4)
  Sore Mouth (Cycle 30/Day 1) (n=107) | -1.2 (12.9)
  Sore Mouth (End of treatment) (n=451) | -0.4 (20.0)

14. Secondary Outcome: Percentage of Participants With Visual Symptom Assessment Questionnaire (VSAQ-ALK)
Description: The participants who responded to the question: "Have you experienced any visual disturbances?" Only the participants who answered yes were instructed to complete the rest of the questionnaire. N was the number of participants who had completed the first question.
Time Frame: 6 years
Population: The safety analysis population included all participants who were enrolled and received at least 1 dose of study medication (excluding day-7 pharmacokinetic [PK] dosing).
Measure: Number; unit: Percentage of participants
Arm/Group | Crizotinib 250 mg BID
Number analyzed (Participants) | 1066
Percentage of participants
  Cycle 2/Day 1 (Yes) (N=798) | 64.5
  Cycle 2/Day 1 (No) (N=798) | 35.5
  Cycle 3/Day 1 (Yes) (N=768) | 56.5
  Cycle 3/Day 1 (No) (N=768) | 43.5
  Cycle 4/Day 1 (Yes) (N=754) | 52.3
  Cycle 4/Day 1 (No) (N=754) | 47.7
  Cycle 5/Day 1 (Yes) (N=743) | 49.1
  Cycle 5/Day 1 (No) (N=743) | 50.9
  Cycle 6/Day 1 (Yes) (N=731) | 48.8
  Cycle 6/Day 1 (No) (N=731) | 51.2
  Cycle 7/Day 1 (Yes) (N=699) | 45.8
  Cycle 7/Day 1 (No) (N=699) | 54.2
  Cycle 8/Day 1 (Yes) (N=670) | 43.7
  Cycle 8/Day 1 (No) (N=670) | 56.3
  Cycle 9/Day 1 (Yes) (N=653) | 43.5
  Cycle 9/Day 1 (No) (N=653) | 56.5
  Cycle 10/Day 1 (Yes) (N=621) | 42.7
  Cycle 10/Day 1 (No) (N=621) | 57.3
  Cycle 11/Day 1 (Yes) (N=565) | 40.2
  Cycle 11/Day 1 (No) (N=565) | 59.8
  Cycle 12/Day 1 (Yes) (N=403) | 42.9
  Cycle 12/Day 1 (No) (N=403) | 57.1
  Cycle 13/Day 1 (Yes) (N=507) | 41.2
  Cycle 13/Day 1 (No) (N=507) | 58.8
  Cycle 14/Day 1 (Yes) (N=354) | 41.5
  Cycle 14/Day 1 (No) (N=354) | 58.5
  Cycle 15/Day 1 (Yes) (N=468) | 39.1
  Cycle 15/Day 1 (No) (N=468) | 60.9
  Cycle 16/Day 1 (Yes) (N=296) | 43.6
  Cycle 16/Day 1 (No) (N=296) | 56.4
  Cycle 17/Day 1 (Yes) (N=418) | 37.3
  Cycle 17/Day 1 (No) (N=418) | 62.7
  Cycle 18/Day 1 (Yes) (N=249) | 40.2
  Cycle 18/Day 1 (No) (N=249) | 59.8
  Cycle 19/Day 1 (Yes) (N=378) | 36.8
  Cycle 19/Day 1 (No) (N=378) | 63.2
  Cycle 20/Day 1 (Yes) (N=221) | 38.9
  Cycle 20/Day 1 (No) (N=221) | 61.1
  Cycle 21/Day 1 (Yes) (N=344) | 39.0
  Cycle 21/Day 1 (No) (N=344) | 61.0
  Cycle 22/Day 1 (Yes) (N=181) | 39.2
  Cycle 22/Day 1 (No) (N=181) | 60.8
  Cycle 23/Day 1 (Yes) (N=312) | 34.9
  Cycle 23/Day 1 (No) (N=312) | 65.1
  Cycle 24/Day 1 (Yes) (N=155) | 34.8
  Cycle 24/Day 1 (No) (N=155) | 65.2
  Cycle 25/Day 1 (Yes) (N=302) | 35.8
  Cycle 25/Day 1 (No) (N=302) | 64.2
  Cycle 26/Day 1 (Yes) (N=130) | 30.8
  Cycle 26/Day 1 (No) (N=130) | 69.2
  Cycle 27/Day 1 (Yes) (N=276) | 32.6
  Cycle 27/Day 1 (No) (N=276) | 67.4
  Cycle 28/Day 1 (Yes) (N=118) | 31.4
  Cycle 28/Day 1 (No) (N=118) | 68.6
  Cycle 29/Day 1 (Yes) (N=249) | 30.5
  Cycle 29/Day 1 (No) (N=249) | 69.5
  Cycle 30/Day 1 (Yes) (N=106) | 27.4
  Cycle 30/Day 1 (No) (N=106) | 72.6
  End of Treatment (Yes) (N=428) | 39.3
  End of Treatment (No) (N=428) | 60.7

15. Secondary Outcome: Patient Reported Outcomes (PROs) of Health-related Quality of Life (HRQoL): Mean Change From Baseline of EQ-5D Visual Analog Score (VAS) Scale
Description: The EQ-5D descriptive system measured a patient's health state on 5 dimensions which included: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The respondent's self-rated health was assessed on a scale from 0 (worst imaginable health state) to 100 (best imaginable health state) by the EQ-VAS. n is the number of participants who completed the scale at baseline and at the respective Cycle.
Time Frame: 6 years
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Crizotinib 250 mg BID
Number analyzed (Participants) | 974
Units on a scale
  CYCLE 2/DAY 1 (n=926) | 5.72 (17.51)
  CYCLE 3/DAY 1 (n=875) | 8.57 (18.82)
  CYCLE 4/DAY 1 (n=836) | 10.01 (19.73)
  CYCLE 5/DAY 1 (n=804) | 10.38 (19.85)
  CYCLE 6/DAY 1 (n=771) | 10.17 (20.38)
  CYCLE 7/DAY 1 (n=728) | 10.17 (20.38)
  CYCLE 8/DAY 1 (n=693) | 10.35 (19.22)
  CYCLE 9/DAY 1 (n=667) | 10.69 (19.82)
  CYCLE 10/DAY 1 (n=633) | 10.34 (19.15)
  CYCLE 11/DAY 1 (n=573) | 10.09 (19.72)
  CYCLE 12/DAY 1 (n=409) | 9.69 (18.81)
  CYCLE 13/DAY 1 (n=512) | 9.74 (19.64)
  CYCLE 14/DAY 1 (n=351) | 10.93 (18.67)
  CYCLE 15/DAY 1 (n=461) | 8.71 (20.53)
  CYCLE 16/DAY 1 (n=289) | 8.47 (20.66)
  CYCLE 17/DAY 1 (n=417) | 7.99 (20.80)
  CYCLE 18/DAY 1 (n=244) | 7.62 (19.86)
  CYCLE 19/DAY 1 (n=372) | 8.17 (18.92)
  CYCLE 20/DAY 1 (n=219) | 8.03 (18.45)
  CYCLE 21/DAY 1 (n=339) | 6.96 (18.71)
  CYCLE 22/DAY 1 (n=179) | 6.59 (18.97)
  CYCLE 23/DAY 1 (n=310) | 5.53 (19.50)
  CYCLE 24/DAY 1 (n=154) | 7.61 (19.58)
  CYCLE 25/DAY 1 (n=299) | 4.97 (17.98)
  CYCLE 26/DAY 1 (n=128) | 8.54 (18.97)
  CYCLE 27/DAY 1 (n=272) | 5.24 (17.61)
  CYCLE 28/DAY 1 (n=120) | 7.93 (19.53)
  CYCLE 29/DAY 1 (n=249) | 5.05 (17.07)
  CYCLE 30/DAY 1 (n=108) | 8.07 (19.95)
  End of Treatment (n=450) | 0.09 (23.92)

16. Primary Outcome: Objective Response Rate
Description: The objective response rate (ORR) as a measure of anti-tumor efficacy of oral PF-02341066 in participants with advanced NSCLC with an ALK gene translocation or inversion after failure of at least one line of chemotherapy.
Time Frame: 6 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Crizotinib 250 mg BID
Number analyzed (Participants) | 1066
Percentage of participants
  ALK Positive by IUO; N=908 | 54.1 [50.8 to 57.4]
  ALK Positive by non-IUO only, N= 158 | 40.5 [32.8 to 48.6]

17. Primary Outcome: Percentage of Participants With Adverse Events
Description: Incidence of adverse events and laboratory abnormalities (severity graded by the National Cancer Institute [NCI] Common Terminology Criteria for Adverse Events [CTCAE], version 4.0).
Time Frame: 6 years
Population: as for outcome 14
Measure: Number; unit: Percentage of Participants
Arm/Group | Crizotinib 250 mg BID
Number analyzed (Participants) | 1066
Percentage of Participants
  Serious AEs (all causalities) | 50.6
  Grade 3/4 AEs (all causalities) | 65.6
  Grade 5 AEs (all causalities) | 22.7
  Serious AEs (treatment related) | 11.5
  Grade 3/4 AEs (treatment related) | 40.2
  Grade 5 AEs (treatment related) | 1.6

ADVERSE EVENTS:
Time Frame: Active reporting period is from the time of informed consent until at least 28 days after study treatment last dose. For serious adverse events: those with the possibility of being related to study drug must be reported as minimum thereafter.
Description: All causality (serious and non-serious) AEs
Arm/Group | Crizotinib 250 mg BID
Serious Adverse Events (participants affected / at risk) | 539/1066
Other Adverse Events (participants affected / at risk) | 1038/1066
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Crizotinib 250 mg BID (N=1066)
Anaemia (Blood and lymphatic system disorders) | 4
Basophilia (Blood and lymphatic system disorders) | 1
Eosinophilia (Blood and lymphatic system disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 6
Leukocytosis (Blood and lymphatic system disorders) | 1
Monocytosis (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Thrombocytosis (Blood and lymphatic system disorders) | 1
Acute myocardial infarction (Cardiac disorders) | 2
Angina pectoris (Cardiac disorders) | 2
Atrial fibrillation (Cardiac disorders) | 3
Bradycardia (Cardiac disorders) | 1
Cardiac arrest (Cardiac disorders) | 2
Cardiac failure (Cardiac disorders) | 2
Cardiac failure congestive (Cardiac disorders) | 1
Cardiac tamponade (Cardiac disorders) | 1
Coronary artery stenosis (Cardiac disorders) | 1
Cyanosis (Cardiac disorders) | 1
Left ventricular failure (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 2
Myocarditis (Cardiac disorders) | 1
Palpitations (Cardiac disorders) | 1
Pericardial effusion (Cardiac disorders) | 7
Pericarditis (Cardiac disorders) | 1
Supraventricular tachycardia (Cardiac disorders) | 1
Syncope (Cardiac disorders) | 6
Tachycardia (Cardiac disorders) | 2
Cataract (Eye disorders) | 2
Glaucoma (Eye disorders) | 1
Optic atrophy (Eye disorders) | 1
Retinal detachment (Eye disorders) | 1
Vision blurred (Eye disorders) | 1
Vitreous haemorrhage (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 6
Abdominal wall haematoma (Gastrointestinal disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 3
Diarrhoea (Gastrointestinal disorders) | 4
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 7
Gastric ulcer (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 3
Ileus (Gastrointestinal disorders) | 3
Intestinal obstruction (Gastrointestinal disorders) | 1
Intestinal perforation (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 9
Oesophageal stenosis (Gastrointestinal disorders) | 1
Oesophagitis (Gastrointestinal disorders) | 2
Pancreatic atrophy (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 3
Pancreatitis acute (Gastrointestinal disorders) | 1
Peptic ulcer haemorrhage (Gastrointestinal disorders) | 1
Peritoneal disorder (Gastrointestinal disorders) | 1
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1
Subileus (Gastrointestinal disorders) | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 6
Asthenia (General disorders) | 7
Chest discomfort (General disorders) | 2
Chest pain (General disorders) | 5
Chills (General disorders) | 1
Condition aggravated (General disorders) | 2
Death (General disorders) | 8
Device dislocation (General disorders) | 1
Disease progression (General disorders) | 135
Fatigue (General disorders) | 4
Gait disturbance (General disorders) | 1
General physical health deterioration (General disorders) | 9
Generalised oedema (General disorders) | 3
Mass (General disorders) | 1
Multi-organ failure (General disorders) | 1
Oedema peripheral (General disorders) | 7
Pain (General disorders) | 1
Pyrexia (General disorders) | 18
Cholecystitis (Hepatobiliary disorders) | 1
Drug-induced liver injury (Hepatobiliary disorders) | 3
Hepatic failure (Hepatobiliary disorders) | 2
Hepatitis (Hepatobiliary disorders) | 1
Hepatocellular injury (Hepatobiliary disorders) | 1
Hepatotoxicity (Hepatobiliary disorders) | 3
Contrast media allergy (Immune system disorders) | 1
Abdominal abscess (Infections and infestations) | 1
Abscess limb (Infections and infestations) | 1
Appendicitis (Infections and infestations) | 8
Bacteraemia (Infections and infestations) | 2
Bone abscess (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 2
Candiduria (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 13
Chest wall abscess (Infections and infestations) | 1
Clostridium difficile infection (Infections and infestations) | 1
Cystitis (Infections and infestations) | 1
Diverticulitis (Infections and infestations) | 1
Empyema (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 6
Herpes zoster (Infections and infestations) | 3
Infection (Infections and infestations) | 1
Infectious pleural effusion (Infections and infestations) | 2
Infective spondylitis (Infections and infestations) | 1
Lower respiratory tract infection (Infections and infestations) | 3
Lung abscess (Infections and infestations) | 1
Lung infection (Infections and infestations) | 14
Meningitis (Infections and infestations) | 1
Metapneumovirus infection (Infections and infestations) | 1
Oesophageal candidiasis (Infections and infestations) | 2
Osteomyelitis chronic (Infections and infestations) | 1
Peritonitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 74
Pneumonia bacterial (Infections and infestations) | 1
Pneumonia fungal (Infections and infestations) | 1
Pneumonia staphylococcal (Infections and infestations) | 1
Pyelonephritis (Infections and infestations) | 1
Renal abscess (Infections and infestations) | 2
Renal cyst infection (Infections and infestations) | 2
Respiratory tract infection (Infections and infestations) | 5
Sepsis (Infections and infestations) | 8
Septic shock (Infections and infestations) | 4
Skin infection (Infections and infestations) | 4
Soft tissue infection (Infections and infestations) | 1
Staphylococcal sepsis (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 7
Urinary tract infection (Infections and infestations) | 7
Urinary tract infection bacterial (Infections and infestations) | 1
Viral infection (Infections and infestations) | 1
Viral upper respiratory tract infection (Infections and infestations) | 1
Wound infection (Infections and infestations) | 2
Ankle fracture (Injury, poisoning and procedural complications) | 2
Bone fissure (Injury, poisoning and procedural complications) | 1
Dislocation of vertebra (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 6
Femoral neck fracture (Injury, poisoning and procedural complications) | 4
Femur fracture (Injury, poisoning and procedural complications) | 4
Hip fracture (Injury, poisoning and procedural complications) | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1
Joint dislocation (Injury, poisoning and procedural complications) | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 1
Overdose (Injury, poisoning and procedural complications) | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 1
Radiation necrosis (Injury, poisoning and procedural complications) | 1
Radiation pneumonitis (Injury, poisoning and procedural complications) | 1
Radius fracture (Injury, poisoning and procedural complications) | 2
Road traffic accident (Injury, poisoning and procedural complications) | 2
Spinal compression fracture (Injury, poisoning and procedural complications) | 2
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1
Traumatic haematoma (Injury, poisoning and procedural complications) | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 5
Blood albumin decreased (Investigations) | 1
Blood bilirubin increased (Investigations) | 1
Blood creatinine increased (Investigations) | 1
Blood lactate dehydrogenase increased (Investigations) | 1
C-reactive protein increased (Investigations) | 1
Electrocardiogram QT prolonged (Investigations) | 1
Hepatic enzyme increased (Investigations) | 1
Troponin I increased (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 3
Dehydration (Metabolism and nutrition disorders) | 4
Failure to thrive (Metabolism and nutrition disorders) | 2
Fluid retention (Metabolism and nutrition disorders) | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 5
Hypomagnesaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 4
Hypophosphataemia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 5
Bursitis (Musculoskeletal and connective tissue disorders) | 1
Chest wall mass (Musculoskeletal and connective tissue disorders) | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Myopathy (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 2
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Pathological fracture (Musculoskeletal and connective tissue disorders) | 5
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Gallbladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Aphasia (Nervous system disorders) | 2
Ataxia (Nervous system disorders) | 1
Brain oedema (Nervous system disorders) | 3
Cerebellar infarction (Nervous system disorders) | 1
Cerebral haemorrhage (Nervous system disorders) | 4
Cerebral infarction (Nervous system disorders) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Chorea (Nervous system disorders) | 1
Coma (Nervous system disorders) | 1
Depressed level of consciousness (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 2
Dysarthria (Nervous system disorders) | 2
Generalised tonic-clonic seizure (Nervous system disorders) | 1
Haemorrhage intracranial (Nervous system disorders) | 1
Headache (Nervous system disorders) | 4
Intracranial pressure increased (Nervous system disorders) | 1
Ischaemic stroke (Nervous system disorders) | 1
Nervous system disorder (Nervous system disorders) | 2
Neurological decompensation (Nervous system disorders) | 1
Paraplegia (Nervous system disorders) | 1
Peripheral motor neuropathy (Nervous system disorders) | 1
Peripheral sensorimotor neuropathy (Nervous system disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1
Pyramidal tract syndrome (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 9
Spinal cord compression (Nervous system disorders) | 2
Transient ischaemic attack (Nervous system disorders) | 3
Tremor (Nervous system disorders) | 1
Vocal cord paralysis (Nervous system disorders) | 2
Completed suicide (Psychiatric disorders) | 1
Confusional state (Psychiatric disorders) | 7
Depression (Psychiatric disorders) | 3
Disorientation (Psychiatric disorders) | 1
Mania (Psychiatric disorders) | 1
Mental status changes (Psychiatric disorders) | 2
Suicide attempt (Psychiatric disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 5
Dysuria (Renal and urinary disorders) | 2
Haematuria (Renal and urinary disorders) | 1
Hydronephrosis (Renal and urinary disorders) | 2
Nephrolithiasis (Renal and urinary disorders) | 2
Renal cyst (Renal and urinary disorders) | 13
Renal cyst haemorrhage (Renal and urinary disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Ureteral polyp (Renal and urinary disorders) | 1
Urinary retention (Renal and urinary disorders) | 2
Urinary tract obstruction (Renal and urinary disorders) | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1
Pelvic pain (Reproductive system and breast disorders) | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3
Alveolitis (Respiratory, thoracic and mediastinal disorders) | 1
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 39
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 4
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 5
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 14
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 4
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 17
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 8
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary artery thrombosis (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 26
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary thrombosis (Respiratory, thoracic and mediastinal disorders) | 1
Rales (Respiratory, thoracic and mediastinal disorders) | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 17
Paraneoplastic pemphigus (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Pleural decortication (Surgical and medical procedures) | 1
Deep vein thrombosis (Vascular disorders) | 14
Embolism (Vascular disorders) | 1
Haematoma (Vascular disorders) | 3
Hypotension (Vascular disorders) | 1
Hypovolaemic shock (Vascular disorders) | 1
Orthostatic hypotension (Vascular disorders) | 1
Peripheral arterial occlusive disease (Vascular disorders) | 1
Peripheral embolism (Vascular disorders) | 2
Phlebitis (Vascular disorders) | 1
Superior vena cava syndrome (Vascular disorders) | 4
Thrombophlebitis (Vascular disorders) | 1
Thrombosis (Vascular disorders) | 5
Vasculitis (Vascular disorders) | 1
Vena cava thrombosis (Vascular disorders) | 2
Venous thrombosis (Vascular disorders) | 4
Angina Unstable (Cardiac disorders) | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1
Vascular stent thrombosis (General disorders) | 1
Lymphangitis (Infections and infestations) | 1
Craniocerebral injury (Injury, poisoning and procedural complications) | 1
Postoperative wound complication (Injury, poisoning and procedural complications) | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 1
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Crizotinib 250 mg BID (N=1066)
Anaemia (Blood and lymphatic system disorders) | 138
Leukopenia (Blood and lymphatic system disorders) | 101
Lymphopenia (Blood and lymphatic system disorders) | 71
Neutropenia (Blood and lymphatic system disorders) | 180
Bradycardia (Cardiac disorders) | 93/1006
Photopsia (Eye disorders) | 96
Vision blurred (Eye disorders) | 80
Visual impairment (Eye disorders) | 460
Abdominal pain (Gastrointestinal disorders) | 118
Abdominal pain upper (Gastrointestinal disorders) | 106
Constipation (Gastrointestinal disorders) | 475
Diarrhoea (Gastrointestinal disorders) | 548
Dyspepsia (Gastrointestinal disorders) | 81
Dysphagia (Gastrointestinal disorders) | 56
Nausea (Gastrointestinal disorders) | 603
Vomiting (Gastrointestinal disorders) | 565
Asthenia (General disorders) | 156
Chest pain (General disorders) | 105
Fatigue (General disorders) | 326
Oedema (General disorders) | 96
Oedema peripheral (General disorders) | 450
Pyrexia (General disorders) | 181
Nasopharyngitis (Infections and infestations) | 113
Upper respiratory tract infection (Infections and infestations) | 145
Urinary tract infection (Infections and infestations) | 62
Fall (Injury, poisoning and procedural complications) | 59
Alanine aminotransferase increased (Investigations) | 302/1006
Aspartate aminotransferase increased (Investigations) | 233/1006
Blood alkaline phosphatase increased (Investigations) | 76/1006
Blood creatinine increased (Investigations) | 105/1006
Blood lactate dehydrogenase increased (Investigations) | 60/1006
Neutrophil count decreased (Investigations) | 84
Weight decreased (Investigations) | 109
Weight increased (Investigations) | 98
White blood cell count decreased (Investigations) | 98/1006
Decreased appetite (Metabolism and nutrition disorders) | 326
Hyperglycaemia (Metabolism and nutrition disorders) | 55
Hypoalbuminaemia (Metabolism and nutrition disorders) | 98
Hypocalcaemia (Metabolism and nutrition disorders) | 99
Hypokalaemia (Metabolism and nutrition disorders) | 77
Arthralgia (Musculoskeletal and connective tissue disorders) | 131
Back pain (Musculoskeletal and connective tissue disorders) | 184
Muscle spasms (Musculoskeletal and connective tissue disorders) | 79
Muscular weakness (Musculoskeletal and connective tissue disorders) | 57
Pain in extremity (Musculoskeletal and connective tissue disorders) | 137
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 74
Dizziness (Nervous system disorders) | 265
Dysgeusia (Nervous system disorders) | 213
Headache (Nervous system disorders) | 214
Hypoaesthesia (Nervous system disorders) | 65
Paraesthesia (Nervous system disorders) | 83
Anxiety (Psychiatric disorders) | 76
Insomnia (Psychiatric disorders) | 136
Cough (Respiratory, thoracic and mediastinal disorders) | 260
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 224
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 55
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 75
Productive cough (Respiratory, thoracic and mediastinal disorders) | 71
Alopecia (Skin and subcutaneous tissue disorders) | 67
Pruritus (Skin and subcutaneous tissue disorders) | 84
Rash (Skin and subcutaneous tissue disorders) | 134
Hyponatraemia (Metabolism and nutrition disorders) | 54

LIMITATIONS AND CAVEATS:
Pharmacogenetic analysis of renal adverse events was not performed as no gene alleles have been identified in published literature with statistically significant association with renal toxicity to support a case control association analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.